# Johnson & Johnson Vision Care, Inc.

## **Clinical Study Protocol**

### Evaluation of Two Marketed Multifocal Contact Lenses

Protocol CR-5860

Version: 3.0, Amendment 2.0

Date: 01-SEP-2017

Investigational Products: Dailies Total 1\* Multifocal Contact Lens and Biotrue ONEday® for Presbyopia Contact Lens.

Key Words: Presbyopia, Daily Disposable, Dispensing, Multifocal, Nesofilcon A, Delefilcon A.

### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP), ISO 14155, the Declaration of Helsinki, and all applicable regulatory requirements.

### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

| | E OF CONTENTS | - |
|---|---|---|
| | OCOL TITLE, NUMBER, VERSION | |
| | SOR NAME AND ADDRESS | |
| | CAL MONITOR | |
| | ORIZED SIGNATURES | |
| CHAN | GE HISTORY | 8 |
| SYNO | PSIS | 9 |
| Figure | 1: Flowchart | 13 |
| COMM | MONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS | 14 |
| 1. IN | FRODUCTION AND BACKGROUND | 16 |
| 1.1. | Name and Descriptions of Investigational Products | 16 |
| 1.2. | Intended Use of Investigational Products | 16 |
| 1.3. | Summary of Findings from Nonclinical Studies | 16 |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | 16 |
| 1.5. | Relevant Literature References and Prior Clinical Data Relevant to Propos Clinical Study | |
| 2. ST | UDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 17 |
| 2.1. | Objectives | 17 |
| 2.2. | Endpoints | 17 |
| 2.3. | Hypotheses | 17 |
| 3. TA | RGETED STUDY POPULATION | 18 |
| 3.1. | General Characteristics | 18 |
| 3.2. | Inclusion Criteria | 18 |
| 3.3. | Exclusion Criteria | 18 |
| 3.4. | Enrollment Strategy | 19 |
| 4. ST | UDY DESIGN AND RATIONALE | 19 |
| 4.1. | Description of Study Design | 19 |
| 4.2. | Study Design Rationale | |
| 4.3. | Enrollment Target and Study Duration | |
| 5. TES | ST ARTICLE ALLOCATION AND MASKING | |
| 5.1. | Test Article Allocation | |
| 5.2. | Masking | |
| 5.3. | Procedures for Maintaining and Breaking Randomization Codes | |
| 6 STI | IDV INTEDVENTION | 21 |

| 6.1. Identity of Test Articles | 21 |
|--------------------------------------------------------|------|
| Table 1: Test Articles | |
| 6.2. Ancillary Supplies/Products | 22 |
| Table 2: Ancillary Supplies | 22 |
| 6.3. Administration of Test Articles | |
| 6.4. Packaging and Labeling | |
| 6.5. Storage Conditions | |
| 6.6. Collection and Storage of Samples | |
| 6.7. Accountability of Test Articles | |
| 7. STUDY EVALUATIONS | |
| 7.1. Time and Event Schedule | |
| Table 3: Time and Events | |
| 7.2. Detailed Study Procedures | |
| VISIT 1 | 28 |
| VISIT 2 | |
| VISIT 3 | 37 |
| VISIT 4 | |
| VISIT 5 | |
| VISIT 6 | |
| FINAL EVALUATION | |
| 7.3. Unscheduled Visits | 50 |
| 7.4. Laboratory Procedures | 51 |
| 8. SUBJECTS COMPLETION/WITHDRAWAL | 52 |
| 8.1. Completion Criteria | 52 |
| 8.2. Withdrawal/Discontinuation from the Study | 52 |
| 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION. | |
| 10. DEVIATIONS FROM THE PROTOCOL | |
| 11. STUDY TERMINATION | |
| 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS. | |
| 13. ADVERSE EVENTS | |
| 13.1. Definitions and Classifications | |
| 13.2. Assessing Adverse Events | 57 |
| 13.2.1 Causality Assessment | 57 |
| 13.2.2 Severity Assessment | , 58 |

| 13.3. | Documentation and Follow-Up of Adverse Events58 | } |
|---|---|---|
| 13.4. | Reporting Adverse Events59 | ) |
| 13 | 3.4.1 Reporting Adverse Events to Sponsor | ) |
| 13 | 3.4.2 Reporting Adverse Events to the Responsible IEC/IRB and Health Author | |
| 13.5. | Event of Special Interest61 | |
| | Reporting of Pregnancy61 | |
| | ATISTICAL METHODS61 | |
| 14.1. | General Considerations61 | |
| | Sample Size Justification61 | |
| | Analysis Populations62 | |
| | Level of Statistical Significance | |
| | Primary Analysis62 | |
| | Secondary Analysis63 | |
| | Other Exploratory Analyses | |
| | Interim Analysis63 | |
| 14.9. | Procedure for Handling Missing Data and Drop-Outs63 | |
| | 2. Procedure for Reporting Deviations from Statistical Plan63 | |
| | TA HANDLING AND RECORD KEEPING/ARCHIVING64 | |
| | Electronic Case Report Form/Data Collection64 | |
| | Subject Record64 | |
| 16. DA | TA MANAGEMENT65 | |
| 16.1. | Access to Source Data/Document65 | |
| 16.2. | Confidentiality of Information65 | |
| 16.3. | Data Quality Assurance65 | |
| 17. MO | NITORING66 | |
| 18. ETI | HICAL AND REGULATORY ASPECTS66 | |
| | Study-Specific Design Considerations | |
| | Investigator Responsibility66 | |
| 18.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB)67 | |
| | Informed Consent68 | |
| | Privacy of Personal Data68 | |
| | JDY RECORD RETENTION69 | |
| | ANCIAL CONSIDERATIONS70 | |

| 21. PUBLICATION70 |
|-----------------------------------------------------------------------------|
| 22. REFERENCES70 |
| APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) 71 |
| APPENDIX B: PATIENT INSTRUCTION GUIDE108 |
| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)109 |
| APPENDIX D: PRESBYOPIC SYMPTOMS QUESTIONNAIRE115 |
| APPENDIX E: OCULAR DOMINANCE116 |
| APPENDIX F: BINOCULAR OVER-REFRACTION117 |
| APPENDIX G: BIOTRUE ONEDAY® FOR PRESBYOPIA FITTING GUIDE118 |
| APPENDIX H: DAILIES TOTAL 1® MULTIFOCAL FITTING GUIDE120 |
| APPENDIX I: CLINICAL TECHNICAL PROCEDURES (CTP)153 |
| , LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS154 |
| , EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING162 |
| DETERMINATION OF NEAR ADD167 |
| NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE175 |
| LENS FITTING CHARACTERISTICS178 |
| SUBJECT REPORTED OCULAR SYMPTOMS185 |
| DETERMINATION OF DISTANCE SPHEROCYLINDRICAL |
| REFRACTIONS |
| BIOMICROSCOPY SCALE |
| KERATOMETRY PROCEDURE |
| , DISTANCE AND NEAR VISUAL ACUITY EVALUATION202 |
| ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE 207 |
| , MEASURING PUPIL DIAMETER WITH NEUROPTICS VIP-200 VARIABLE PUPILLOMETER211 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE215 |
| A TOTALIC OF TABLES |
| LISTING OF TABLES |
| Table 1: Test Articles |
| Table 3: Time and Events |
| LISTING OF FIGURES |
| Figure 1: Flowchart |

### PROTOCOL TITLE, NUMBER, VERSION

Title: Evaluation of Two Marketed Multifocal Contact Lenses

Protocol Number: CR-5860 Version: 3.0, Amendment 2.0

Date: 01-SEP-2017

### **SPONSOR NAME AND ADDRESS**

Johnson & Johnson Vision Care, Inc. (JJVC) 7500 Centurion Parkway, Jacksonville, FL 32256

### **MEDICAL MONITOR**

NAME: Thomas R. Karkkainen, OD, MS, FAAO

TITLE: Sr. Principal Research Optometrist

ADDRESS: 7500 Centurion Parkway, Jacksonville, Florida 32256

E-MAIL: TKarkkai@its.jnj.com

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

### **AUTHORIZED SIGNATURES**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations, ICH guidelines, ISO 14155 and the Declaration of Helsinki.

| Author | | |
|---|---|---|
| | Thomas R. Karkkainen, OD, MS, FAAO<br>Title: Sr. Principal Research Optometrist | DATE |
| Clinical Operations<br>Manager | | |
| | Clinical Operations Manager | DATE |
| Biostatistician | | |
| | Biostatistician IV | DATE |
| Data Management | | |
| | Clinical Project Manager-Data and<br>Systems | DATE |
| Approver | | |
| <del>.</del> | Presbyopia Platform Sr. Manager | DATE |

### **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section<br>Number(s) Affected | Date |
|---|---|---|---|
| 1.0 | Tom Karkkainen | Original Protocol | 23-June-2017 |
| 2.0 | | Change Secondary Objective on page 17 to CLUE vision score. | 30-June-2017 |
| 3.0 | Tom Karkkainen | In section 2.3 updated hypotheses. | 01-September-<br>2017 |

### **SYNOPSIS**

| Protocol Title | Evaluation of Two Marketed Multifocal Contact Lenses |
|---|---|
| Sponsor JJVC, 7500 Centurion Parkway, Jacksonville, FL 322 | |
| Clinical Phase | Development phase, phase 0 (Research) |
| Trial Registration | This study will be registered on ClinicalTrials.gov by the Sponsor |
| Test Article(s) | Investigational Products: Biotrue ONEday and Oneday for Presbyopia and Dailies Total 1 Multifocal Contact Lenses. Control Products: None |
| Wear and Replacement | Wear Schedule: Daily |
| Schedules | Replacement Schedule: Daily Disposable |
| Objectives | Primary Objective: |
| | To evaluate the visual performance of a marketed multifocal contact lens in a population of presbyopes with myopia and hyperopia. |
| | Secondary Objective: |
| | CLUE vision score |
| Study Endpoints | Primary endpoints: The primary endpoints in this study are distance and near binocular high luminance, high contrast visual performance on logMAR scale. |
| | Secondary endpoint: The secondary endpoint is overall quality of vision assessed using the Contact Lens User Evaluation questionnaire (CLUE <sup>TM</sup> ). |
| | Other endpoint: Ease of fit as evaluated by the number of lenses used to optimize. |

| Study Design Sample Size | This is a single-masked, randomized, cross-over, dispensing pilot study. There will be six study visits. Visit 1 will include baseline measurements and screening to ensure eligibility. Eligible subjects will be randomized and fit in one of the study lenses and dispensed for 2-4 days. At Visit 2 additional measurements will be performed and it will be determined if lens optimization is required and lenses dispensed for an additional 6-8 days. At Visit 3 the primary endpoint data used for analysis will be collected. There will be a 4-8-day washout before the subject will be fit with the 2 <sup>nd</sup> lens at Visit 4 and dispensed for 2-4 days. At Visit 5 additional measurements will be performed and it will be determined if lens optimization is required and lenses dispensed for an additional 6-8 days. At Visit 6 the primary endpoint data used for analysis will be collected. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations. A total of approximately 80 eligible subjects will be enrolled into the study with 60 (30 myopes and 30 hyperopes) subjects targeted to complete the study. An attempt will be made to evenly distribute the subjects across the following ADD | |
|---|---|---|
| | evenly distribute the subjects across the following ADD groups. | |
| | ADD 0.75 D to 1.50 D | ADD 1.75 D to 2.50 D |
| | 30 Subjects | 30 Subjects |
| Study Duration | The study recruitment is anticipated to be approximately 3 weeks and the data collection approximately and additional 3 weeks. | |
| Anticipated Study | Habitual contact lens wearer who are myopic or hyperopic and | |
| Population | have presbyopia. | |
| Eligibility Criteria | Potential subjects must satisfy all | of the following criteria to |
| | be enrolled in the study: 1. The subject must read, under | stand and sion the |
| | 1 | ED CONSENT and receive a |
| | fully executed copy of the for | |
| | 2. The subject must appear able | • |
| | instructions set forth in this c | • |
| | 3. The subject must be between | • |
| | not greater than 70 years of age. 4. The subject's distance spherical equivalent refraction be in the range of +3.75 D to -3.75 D. | |

- 5. The subject's refractive cylinder must be  $\leq$  -0.75 D in each eye.
- 6. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.
- 7. The subject must have best corrected visual acuity of  $20/20^{-3}$  or better in each eye.
- 8. The subject must own a pair of wearable spectacles if required for their distance vision.
- 9. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month or more duration).
- 10. The subject must either be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Ocular or systemic allergies or disease, or use of medication which might interfere with contact lens wear.
- 2. Pregnancy or lactation.
- 3. Currently diagnosed with diabetes.
- 4. Infectious diseases (e.g. hepatitis, tuberculosis) or an immune-suppressive disease (e.g. HIV).
- 5. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
- 6. Entropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
- 7. Any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
- 8. A history of amblyopia, strabismus or binocular vision abnormality.
- 9. Any ocular infection or inflammation.
- 10. Any ocular abnormality that may interfere with contact lens wear.
- 11. Use of any ocular medication, with the exception of rewetting drops.
- 12. History of herpetic keratitis.
- 13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.

| | 14. Employee of clinical site (e.g., Investigator, Coordinator, Technician) |
|---|---|
| Disallowed | Any systemic medications that may affect contact lens wear |
| Medications/Interventions | and any ocular medications with the exception of rewetting |
| | drops. Previous ocular or intraocular surgery. |
| Measurements and | The key assessments for this study will be distance and near |
| Procedures | binocular high luminance, high contrast visual performance on |
| | logMAR scale and overall quality of vision assessed using the |
| | Contact Lens User Evaluation questionnaire (CLUE <sup>TM</sup> ). |
| Microbiology or Other | None |
| Laboratory Testing | |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device |
| | Effect (UADE), or any SAE where relationship to study agent |
| | cannot be ruled out, will result in stopping further dispensing |
| | investigational product. In the event of a UADE or SAE, the |
| | Sponsor Medical Monitor may unmask the treatment regimen |
| | of subject(s) and may discuss this with the Principal |
| | Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study- | ETDRS light box and logMAR High Contrast and Low |
| Specific Materials | Contrast 3M charts, Guillon-Poling Near Charts, Desk lamps, |
| | Chart holder, Sekonic light meter, Pupillometer, Contact lens |
| | cases, and Eye-Cept® rewetting drops. |
| Principal Investigator(s) | A full list of Principal Investigators, clinical sites, and |
| and Study | institutions is kept separately from the Study Protocol and is |
| Institution(s)/Site(s) | included in the study Trial Master File. |

Figure 1: Flowchart



### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required for Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience

BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

CLDEQ-8 8-Item Contact Lens Dry Eye Questionnaire COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

CTP Clinical Technical Procedure

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDEInvestigational Device ExemptionIECIndependent Ethics CommitteeIRBInstitutional Review BoardIRTItem Response Theory

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution MedDRA® Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye
OU Both Eyes

PD Protocol Deviation

| PHI | Protected Health Information |
|-----|------------------------------|

PI Principal Investigator
PIG Patient Instruction Guide
PQC Product Quality Complaint
PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

### 1. INTRODUCTION AND BACKGROUND

Johnson & Johnson Vision recently launched a daily disposable multifocal contact lens, 1-Day ACUVUE® Brand MOIST® Multifocal. Since the launch of this lens additional daily disposable multifocal contact lenses have been approved and marketed. The purpose of this clinical study is to evaluate the performance of two of the newer competitor lenses that have been launched. The data will help to better understand the performance strengths and weaknesses of each product.

### 1.1. Name and Descriptions of Investigational Products

This study will test two (2) marketed multifocal contact lenses, Biotrue ONEday<sup>®</sup> for Presbyopia and Dailies Total 1<sup>®</sup> Multifocal Contact Lens. Further details about the test articles are found in Section 6 of this protocol.

### 1.2. Intended Use of Investigational Products

The intended use of the lenses is to correct distance spherical refractive error and presbyopia. Greater details on each of the marketed products can be found in the package insert in the appendices of this protocol.

### 1.3. Summary of Findings from Nonclinical Studies

Not Applicable – Marketed product only.

### 1.4. Summary of Known Risks and Benefits to Human Subjects

The contact lenses are currently marketed products that, like all multifocal contact lenses, act as a refractive media to correct for distance spherical refractive error and presbyopia. Beyond having their vision corrected by the contact lenses the subject will have no direct benefit from participating in the study.

The intent of these products is for use as a daily disposable contact lens that the subject wears while awake. The lenses are not intended for extended wear or reuse. This evaluation is for daily disposable modality only. Anticipated risks and adverse reactions with this lens are like other soft daily wear contact lenses used to correct presbyopia. A listing of examples of adverse reactions is found in the Section 13 of this protocol. The Investigator should follow normal clinical guidelines regarding examination and care of subjects who participate in this trial. For the most comprehensive clinical information regarding the marketed products refer to the package insert for the marketed product locate in the appendices of this clinical protocol.

### 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

A PubMed literature search using the term "Biotrue Oneday for Presbyopia" and "Dailies Total 1 Multifocal Contact Lens" revealed no results. Additional information regarding the marketed products can be found in the package inserts located in the appendices of this clinical protocol.


### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

### 2.1. Objectives

### **Primary Objective:**

To evaluate the visual performance of a marketed multifocal contact lens in a population of presbyopes with myopia and hyperopia.

### Secondary Objective:

CLUE vision score

Exploratory Objective: Not Applicable

### 2.2. Endpoints

### **Primary Endpoint**

The primary endpoint in this study are distance and near binocular high luminance, high contrast visual performance on logMAR scale.

### Secondary Endpoint

The secondary endpoint is overall quality of vision assessed using the Contact Lens User Evaluation questionnaire (CLUE<sup>TM</sup>). CLUE is a validated Patient Reported Outcome (PRO) questionnaire developed to measure general and throughout the day comfort/vision, as well as symptoms of discomfort/poor vision, lens handling and packaging. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. A 5-point increase in an average CLUE score translates into 10% shift in the distribution of scores for population of soft contact lens wearers. Both primary and secondary endpoints will be assessed after wearing each optimized study lens for 6-8 days.

### Other Observations:

The other endpoints are the ease of fit as measured by the total number of lenses required to optimize vision each lens type and the ocular physiological response are measured by the average corneal staining grade using the FDA biomicroscopy scale for corneal staining. The data for the ease of fit and corneal staining will be summarized.

### 2.3. Hypotheses

### **Primary Hypotheses**

- 1. After 8-12 days of lens wear, the distance, binocular, high luminance, high contrast visual performance of the two test lenses will be superior to +0.01 logMAR.
- 2. After 8-12 days of lens wear, the near, binocular, high luminance, high contrast visual performance of the two test lenses will be superior to +0.17 logMAR.

### Secondary Hypothesis

1. After 8-12 days of lens wear, the overall quality of vision of the two test lenses will be superior to 32 CLUE points.

Other Hypotheses: Not applicable.

### 3. TARGETED STUDY POPULATION

### 3.1. General Characteristics

Healthy male and female volunteers who are presbyopic will be recruited for the study. The subjects will all be adapted wearers of soft contact lenses in both eyes.

### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. The subject must be between at least 40 years of age and not greater than 70 years of age.
- 4. The subject's distance spherical equivalent refraction must be in the range of +3.75 D to -3.75 D.
- 5. The subject's refractive cylinder must be  $\leq$  -0.75 D in each eye.
- 6. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.
- 7. The subject must have best corrected visual acuity of 20/20<sup>-3</sup> or better in each eye.
- 8. The subject must own a pair of wearable spectacles if required for their distance vision.
- 9. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month or more duration).
- 10. The subject must either be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Ocular or systemic allergies or disease, or use of medication which might interfere with contact lens wear.
- 2. Pregnancy or lactation.
- 3. Currently diagnosed with diabetes.
- 4. Infectious diseases (e.g. hepatitis, tuberculosis) or an immune-suppressive disease (e.g. HIV).
- 5. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
- 6. Entropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
- 7. Any previous, or planned, ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
- 8. A history of amblyopia, strabismus or binocular vision abnormality.
- 9. Any ocular infection or inflammation.

- 10. Any ocular abnormality that may interfere with contact lens wear.
- 11. Use of any ocular medication, with the exception of rewetting drops.
- 12. History of herpetic keratitis.
- 13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 14. Employee of clinical site (e.g., Investigator, Coordinator, Technician)

### 3.4. Enrollment Strategy

Study subjects will be recruited from the clinical site's subject database.

### 4. STUDY DESIGN AND RATIONALE

### 4.1. Description of Study Design

This is a single-masked, crossover, randomized, dispensing clinical trial. A total of approximately 60 eligible subjects will be targeted to complete the study. The subjects will be randomized and fit in the study lens and wear each lens type for approximately three days then undergo optimization, if required, and wear the optimized pair for approximately 1 week. The primary endpoint is visual performance. The secondary endpoint is the CLUE vision score.

### 4.2. Study Design Rationale

The study is a prospective, bilateral, crossover evaluation. As we have no historical clinical data on the lenses being tested the study design includes a washout period to minimize any potential carry-over effect.

### 4.3. Enrollment Target and Study Duration

Approximately 80 subjects will be recruited (40 myopes and 40 hyperopes) with an aim of completing a total of 60 subjects in the final cohort.

### 5. TEST ARTICLE ALLOCATION AND MASKING

### 5.1. Test Article Allocation

The study lenses will be worn in a bilateral and random fashion using a 2×2 crossover design with 2 lens types and 2 periods. Using a computer-generated randomization scheme provided by the study biostatistician, each subject will randomly be assigned to one of two unique sequences of the two lens types (Test1/Test2 or Test2/Test1). Randomization will be stratified by site.

Permuted block randomization will be used to avoid bias in the assignment of subjects to treatment, and to enhance the validity of statistical comparisons across treatment groups. Each block will contain two different lens trial sequences.

The order of lens wear will be based on the randomization scheme assigned to the study site. The study site will follow the randomization scheme provided and will complete enrollment according to the randomization list and will not pre-select or assign subjects.

This is a single masked study: subjects will be masked to the identities of the study lenses.

### 5.2. Masking

Masking will be used to reduce potential bias. Subjects will be unaware of the identity of the investigational product. Investigators and clinical site personnel involved in the data collection will not be masked as to the identity of the investigational product.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken; the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

### 5.3. Procedures for Maintaining and Breaking Randomization Codes

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme.
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section

### 6. STUDY INTERVENTION

### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Test 1 | Te | st 2 |
|---|---|---|---|
| Name | Dailies Total 1® | Biotrue ONEday® | Biotrue ONEday® |
| | Multifocal | for Presbyopia | Contact Lenses |
| | Contact Lens | Contact Lens | |
| Manufacturer | Alcon® | Bausch and Lomb | Bausch and Lomb |
| Compass Protocol(s) and/or Lot | Over-labeled | Over-labeled | Over-labeled |
| Number or Other Identifier | | | |
| Lens Material | delefilcon A | nesofilcon A | nesofilcon A |
| Nominal Base Curve @ 22°C | 8.5 | 8.6 | 8.6 |
| Nominal Diameter @ 22°C | 14.1 | 14.2 | 14.2 |
| Nominal Distance Powers (D) | +4.25 D | +4.50 D to -4.00 | +4.00 D to -4.00 |
| | to -4.00 D | D in 0.25 D steps | D in 0.25 D steps |
| | in 0.25D steps | | |
| Nominal ADD Powers (D) | LO | Low | Not Applicable |
| | MED | (+0.75 to +1.50 | |
| | HI | Spectacle Add) | |
| | | High | |
| | | (+1.75 to +2.50 | |
| | | Spectacle Add) | |
| Water Content | 33% (Core | 78% | 78% |
| | Water Content) | | |
| Center Thickness | 0.09 mm | 0.1 mm (-3.00 D) | 0.1 mm (-3.00 D) |
| | (-1.00 D) | | |
| Oxygen Permeability (Dk) | 156 @ -3.00D | 42 @center for | 42 @center for |
| | | -3.00 D | -3.00D |
| Modality in Current Study | Daily | Daily Disposable | Daily Disposable |
| | Disposable | | |
| Replacement Frequency | Daily | Daily | Daily |
| Packaging Form (vial, blister, | Blister | Blister | Blister |
| etc.) | | | |

Each subject what completes the study will wear approximately 22 lenses. As there are 60 subjects approximately 1320 lenses would be used for each lens type.

### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Solution |
|---------------------------|---------------------------|
| Solution Name/Description | Eye-Cept® Rewetting drops |
| Manufacturer | Optics Laboratory |
| Preservative | Non-preserved |

### 6.3. Administration of Test Articles

Test articles will be dispensed to subject meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

### 6.4. Packaging and Labeling

The test articles will be packaged in blisters, as the primary packaging. The test article will be over-labeled to mask the subject to the identity of the lens. The test articles will be in investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study label is shown below:



### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

### 6.6. Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJVC.

### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits
- 2. What was returned to the Investigator unused
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles, and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will package and return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately.</u>

# 7. STUDY EVALUATIONS

# 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 |
|---|---|---|---|---|---|---|
| | Screening, Baseline, Treatment 1 | Treatment 1<br>Follow-up 1 | Treatment 1<br>Follow-up 2 | Baseline 2<br>Treatment 2 | Treatment 2 Follow-up 1 | Treatment 2 Follow-up 2 Final Evaluation |
| Fime Point | Day 1 | Day 3±1 from<br>VI | Day 7±1 from<br>V2 | Day 6±2 from<br>V3 | Day 3±1 from V4 | Day 7±1 from V5 |
| Estimated Visit Duration | 2.5 hours | 1.5 hours | 1.5 hours | 1.5 hours | 1.5 hours | 1.5 hours |
| Statement of<br>Informed Consent | X | | | | | |
| Demographics | × | | | | | |
| Medical<br>History/Concomitant<br>Medications | × | | | | | |
| Adverse Event<br>Medical<br>History/Concomitant<br>Medications Review | | × | × | × | × | × |
| Habitual Contact<br>Lens Information | X | | | | | |
| Contact Lens<br>History | X | | | | | |
| Wear Time | X | X | X | | × | X |
| Screening<br>Inclusion/Exclusion | × | | | | | |

| Visit 6 Treatment 2 Follow-up 2 Final Evaluation | Day 7±1 from V5 | 1.5 hours | | | X | × | × | × | | × | | | X | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day 3±1 from V4 Da | 1.5 hours | | | X | X | × | X | | Х | | | X | | | | | |
| | Day 6±2 from Day V3 | 1.5 hours | | × | x | x | | X | | × | | | X | | | | | |
| Visit 3 Treatment 1 Follow-up 2 | Day 7±1 from<br>V2 | 1.5 hours | | | x | X | X | × | | x | | | x | | | : | | |
| Visit 2<br>Treatment 1<br>Follow-up 1 | Day 3±1 from V1 | 1.5 hours | | | × | X | X | × | | X | | | X | | | | | - |
| Visit 1 Screening, Baseline, Treatment 1 | Day 1 | 2.5 hours | | × | × | | | X | X | × | | × | X | X | X | X | Х | × |
| Visit Information | Time Point | Estimated Visit Duration | Criteria | Baseline PRO<br>Ouestionnaire | CIDEQ-8<br>Ouestionnaire | PRO Questionnaire | Compliance | Subject Reported<br>Ocular Symptoms | Screening Eligibility | Entrance Snellen<br>Distance Visual | Acuty | Subjective Sphero-<br>Cylindrical<br>Refraction | Lens Removal | Pupillometry | Keratometry | Near Add<br>Determination | Ocular Dominance | Add Refinement |

| o<br>ent 2<br>up 2<br>luation | rom V5 | UITS | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Visit o Treatment 2 Follow-up 2 Final Evaluation | Day 7±1 from V5 | 1.5 hours | | 7 | | | | X |
| Visit 5<br>Treatment 2<br>Follow-up 1 | Day 3±1 from V4 | 1.5 hours | | × | × | × | × | |
| V<br>Trea<br>Foll | Day 34 | 77 | | | | | | |
| Visit 4 Baseline 2 Treatment 2 | Day 6±2 from<br>V3 | 1.5 hours | | × | × | × | × | |
| V.<br>Bas:<br>Trea | | 1.5 | | | | | | |
| Visit 3 Treatment 1 Follow-up 2 | Day 7±1 from<br>V2 | 1.5 hours | | | × | | X | |
| | | | | | | - | | |
| Visit 2 Treatment 1 Follow-up 1 | Day 3±1 from<br>VI | 1.5 hours | | X | X | × | X | |
| t.1<br>ing,<br>ine,<br>ent.1 | | SILLS | | | | | | |
| Visit 1 Screening, Baseline, Treatment 1 | Day 1 | 2.5 hours | | X | X | × | × | |
| ion | 1 | it. | (if | riteria | | | dn-mo | ion |
| Visit Information | Time Point | Estimated Visit<br>Duration | Unworn Lens (if applicable) | Dispensing Criteria | Instructions | Dispense Test<br>Article | Schedule Follow-up | Final Evaluation |
| Visi | Tim | Esti.<br>Der | Unv | Dist | Inst | Disj. | Sch | Fin |

### 7.2. Detailed Study Procedures

### VISIT 1

Subjects must report to the visit wearing their habitual contact lenses, to accurately assess baseline CLUE performance. If the subject is not wearing their lenses they must be rescheduled.

| | | Visit 1: Screening | |
|---|---|---|---|
| Step | Procedure | Details | 111 |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign<br>the Statement of Informed Consent before<br>being enrolled into the study. The Principal<br>Investigator or his/her designee conducting<br>the informed consent discussion must also<br>sign the consent form. | |
| | | Note: The subject must be provided a signed copy of this document. | |
| 1.2 | Demographics | Record the subject's date of birth, gender, race and ethnicity. | |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. | |
| 1.4 | Habitual Lenses | Record the brand of their current contact lens, lens parameters, modality (i.e. daily wear, extended wear, etc.) and cleaning regiment. | |
| 1.5 | Contact Lens<br>History | Record the subject's correction type (i.e. monovision, multifocal, sphere with readers, etc.). | |
| 1.6 | Wear Time | Record the subjects wear time and comfortable wear time with their habitual contact lenses. | |
| 1.7 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. | |

| | and the second | Visit 1: Baseline |
|---|---|---|
| Step | Procedure | Details |
| 1.8 | Baseline Questionnaire and CLDEQ-8 Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of their habitual lenses using the PRO questions and the Contact Lens Dry Eye Questionnaire |

| 1.9 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
|---|---|---|---|
| 1.10 | Entrance Distance<br>and Near Visual<br>Acuity | Record the distance and near Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual contact lens correction in place. | |
| | | For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| 1.11 | Lens Removal | Have the subject remove their habitual lenses and store in an approved solution. | |
| 1.12 | Pupillometry | The pupil measurements will be performed OD and OS under bright illumination (7.3-7.9 EV) and dark illumination (≤0 EV) using a Neuroptic Pupillometer or similar instrument. The room illuminance will be measured for each condition using the Sekonic lightmeter or similar instrument. | |
| 1.13 | Keratometry | Keratometry will be performed OD and OS recording the steep and flat dioptric power, corresponding meridians and clarity of mires. | |
| 1.14 | Subjective Sphero-<br>cylindrical<br>Refraction | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. Record the refraction and distance visual acuity to the nearest letter. Note: Best distance visual acuity with | |
| | | sphero-cylindrical refraction must be at least $20/20^{-3}$ in each eye for the subject to enroll in the study. | |
| 1.15 | Near ADD<br>Determination | The near reading addition will be determined using the binocular crossed cylinder technique at 40 cm followed by optimization in a trial frame in step 1.17 below. | |
| 1.16 | Ocular Dominance | Determine the distance ocular dominance with the best distance correction in place using a +1.00-blur test. If the results are equivocal use the sighting dominance test to determine the dominant eye used for the study | Appendix E |
| 1.17 | Add Refinement | Place the BCC result in the trial frame and refine the near prescription with trial lenses (or flippers) under binocular conditions. | |
| 1.18 | Near Visual Acuity | Using the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm. Record the near visual acuity OD, OS and OU at 40 cm. | |

| 1.19 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. For the conjunctival redness ( ) 0.5 unit increments will be used in the grading. Corneal Staining Assessment ( |
|---|---|---|
| | | will be graded in 1.0 increments. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 1.20 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. |
| | | Determine whether the subject is eligible to participate in the study based on the examination findings. If so, proceed to lens fitting. If not, complete the final evaluation and discharge the subject. |

| | 24796 J | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.21 | Randomization ID | Record the Randomization ID per the random scheme. | |
| 1.22 | Lens Selection | Select the lens pair and power based on the randomization table and appropriate fitting guide for each eye. Record the test lens parameters (power and lot number). | Appendix G or H Fitting |
| | | | Guides |
| 1.23 | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. | |
| - | | Check for lens damage under the slit lamp<br>before proceeding with lens settling. | |
| | | Replace damaged lenses if applicable. Worn, damaged lenses must be saved in saline and a product complaint form | |
| 1.24 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. | |
| 1.25 | Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look | |

| | | 1 1 11 2 2 4 4 2 | |
|---|---|---|---|
| | | down a hallway or out of a window for | |
| | | distance vision assessments, and for them to | |
| | | read a book, magazine or similar for near | |
| | | vision. | |
| 1.26 | Distance and Near | Measure the distance and near visual acuity | |
| | Visual Acuity | OD, OS and OU. Record the results. | |
| | | Note: Use the ETDRS 2000 Series Chart 1 or | |
| | | 2 near card placed at 40 cm to measure the | |
| | | Near visual acuity | |
| 1.27 | Over-refraction | Perform a distance over-refraction OD and | |
| 1.27 | Over-remaction | OS using loose lenses outside of the | |
| | | phoropter under ambient room illumination. | |
| | | 1 = " | |
| | | The distance over-refraction may also be | |
| | | refined under binocular conditions. Record | |
| | | the results. | |
| | | The woulder of the distance of the | |
| | | The results of the distance over-refraction | |
| | | may also be checked for the impact on near | |
| | | vision under monocular and/or binocular | |
| 1.00 | | conditions. | |
| 1.28 | Lens Fit | Evaluate and grade lens centration, primary | |
| | Assessment | gaze movement, upgaze movement and | |
| | | tightness (push-up test). | |
| | | The subject will not proceed to wear the | |
| | | lenses if any of the following is observed: | |
| | | <ul> <li>presence of limbal exposure</li> </ul> | |
| | | (appearance of clear cornea) in any | |
| | | gaze | |
| | | <ul> <li>presence of edge lift</li> </ul> | |
| | | presence of unacceptable movement | |
| | | (excessive or insufficient) in all three | |
| | | movement categories (primary gaze, | |
| | | upgaze, and push-up). | |
| | | upgaze, and pash up). | |
| | | If either lens is deemed unacceptable, the | |
| | | subject will be discontinued from the study. | |
| | | Remove the lenses, perform a slit-lamp | |
| | | evaluation, and complete the Final | |
| 1.20 | Madifications | Evaluation form. | A mm arr -11 |
| 1.29 | Modifications | If the subjects vision is unacceptable for at | Appendix |
| | | least one distance or the Investigator | G or H |
| | | determines that the visual acuity or over- | |
| | | refraction are not acceptable then a lens | Fitting |
| | | modification must be made. | Guides |
| | | Up to two attempts at modification are | |

| | | permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the appropriate fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. If modifications are required steps 1.22-1.28 will be repeated for each modification. |
|---|---|---|
| 1.30 | PRO Post-Fit<br>Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire. |
| 1.31 | Exit Distance and<br>Near Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. Note: The distance visual acuity must be at |
| 1.32 | Dispensing<br>Criteria | least 20/30 OU for the lenses to be dispensed. The lenses will be dispensed for 2-4 days. Distance Snellen acuity equal to or better than 20/30 OU Subject must indicate that the vision is acceptable. Subject must indicate that the comfort of the lenses is acceptable. Lenses must have an acceptable general lens fit. |
| 1.33 | Subject<br>Instructions | Instruct the Subject the following: • The lenses will be worn on a daily wear basis. • Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed. • A new lens will be opened and worn each day. • Instruct the subject to bring back all Unworn study lenses • Instruct the subject no cleaning or |

| | | disinfecting solutions will be used. If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness. Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study. Subjects will be instructed to wear their glasses when not wearing the study lenses. A patient instruction booklet will be provided. |
|---|---|---|
| | | Note: In the event a lens is lost or damaged, the subject will return to the clinical site for |
| | | replacement. As much as reasonably |
| i . | | possible, a damaged lens and packaging |
| | : | should be returned to the clinical site (wet, if |
| | | possible) and then returned to the Sponsor. If lens damage is present, complete the Product |
| | · | Quality Complaint Form. The lens will be |
| | | stored in labeled vial with saline, and clearly |
| | | differentiated from the other worn lenses that |
| | | will be shipped back to the Sponsor. |
| 1.34 | Schedule Follow-up | The subject will be scheduled to return for |
| | Visit | their follow-up appointment in 3±1 days. |
| | | Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

### VISIT 2

The subjects must present to Visit 2 wearing the study lenses.

| | Visit 2: Treatment 1 Follow-Up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 2.1. | Adverse Events,<br>Medical History and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 2.2. | Wearing Time | Record the average wearing time and comfortable wearing time. |
| 2.3. | Compliance | Confirm compliance with the prescribed wear schedule. |

| | | | 7 |
|---|---|---|---|
| | | Note: Subjects must have worn lenses for at least 6 hours per day. To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. | |
| 2.4. | PRO and CLDEQ-8 Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire and the Contact Lens Dry Eye Questionnaire | |
| 2.5. | Subject Reported Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 2.6. | Visual<br>Satisfaction | Record whether the subjects distance and near vision with the lenses is acceptable. | |
| 2.7. | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU to the nearest letter. Record the results. | |
| | | Note: Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity | |
| 2.8. | Distance Over-<br>refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results and distance visual acuity OD and OS. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 2.9. | Determination of Lens Optimization | If the subjects vision is unacceptable for at least one distance or the Investigator determines that the visual acuity or overrefraction are not acceptable then a lens modification must be made. Up to two attempts at modification are permitted if necessary, to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that lens type. Follow the appropriate fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. | Appendix G or H Fitting Guides |

| 2.10. | Lens Fit | Evaluate and grade lens centration, primary | |
|---|---|---|---|
| | Assessment | gaze movement, upgaze movement and | |
| | | tightness (push-up test). | |
| | | The subject should not proceed to | |
| | | wear the lenses if any of the following | |
| | | is observed: | |
| | | <ul> <li>presence of limbal exposure</li> </ul> | |
| | | (appearance of clear cornea) in any | |
| | | gaze | |
| | | <ul> <li>presence of edge lift</li> </ul> | |
| | | <ul> <li>presence of unacceptable movement</li> </ul> | |
| | | (excessive or insufficient) in all three | |
| | | movement categories (primary gaze, | |
| | | upgaze, and push-up). | |
| | | If either lens is deemed unacceptable, the | |
| | | subject will be discontinued from the study. | |
| | | Remove the lenses, perform a slit-lamp | ļ |
| | | evaluation, and complete the Final Evaluation | |
| | | form. | |
| 2.11. | Collection of | Collect unworn lenses returned by the subject | |
| : | unworn lenses | when lens power has been optimized. | |
| | | Note: If lens power was not changed allow the | |
| | | subject to use the unworn lenses dispensed at | |
| | | Visit 1 and dispense enough lenses of the | |
| | | same power to last the subject until their next | |
| | 1 | visit. | |
| 2.12. | Lens Removal | The optimized study lenses will be removed | |
| 2.12 | Diamiaragaany | and discarded. FDA Slit Lamp Classification Scale will be | |
| 2.13. | Biomicroscopy | used to grade the findings and determine | |
| | | eligibility. | |
| | | For the conjunctival redness 0.5 | |
| | | unit increments will be used in the grading. | |
| | | Corneal Staining Assessment will | |
| | | be graded in 1.0 increments. | |
| | | If the clearance of the fluorescein needs to be | |
| | | expedited, preservative-free rewetting drops | |
| | | or saline may be instilled. | |
| 2.14. | Insertion of Study | Dispense the subject new lenses that match | |
| 2.17. | Lenses | the Distance and ADD power of the lenses | |
| | | that were removed in Step 2.12 above. | |
| | | Dispense enough lenses to last the subject | |
| | | 2.50 | <del></del> |

| | <del></del> | |
|---|---|---|
| | | until their next visit. |
| 2.15. | PRO Questionnaire | The subject will evaluate the vision |
| | | characteristics, comfort characteristics, |
| | | handling characteristics, and visual symptoms |
| | | of the study lenses using the PRO |
| | | questionnaire. |
| 2.16. | Exit Distance and | Distance and near Snellen visual acuity will |
| | Near Visual Acuity | be measured for each eye with the study |
| | | contact lenses in place. |
| | | For near measures use the ETDRS 2000 |
| | | Series Chart 1 or 2. The acuity will be |
| | | recorded to the nearest letter OD, OS and OU. |
| 2.17. | Dispensing | The lenses will be dispensed for 6-8 days. |
| 2.17. | Criteria | |
| | Cittoria | Distance Snellen acuity equal to or hotten them 20/20 OII. |
| | | better than 20/30 OU |
| | | Subject must indicate that the vision is |
| | | acceptable. |
| | | Subject must indicate that the comfort |
| | | of the lenses is acceptable. |
| | | • Lenses must have an acceptable |
| - 1 i | | general lens fit. |
| 2.18. | Subject | Instruct the Subject the following: |
| | Instructions | • The lenses will be worn on a daily |
| | | wear basis. |
| | | <ul> <li>Only enough lenses will be dispensed</li> </ul> |
| | | to the subject to wear for the required |
| | | number of days until their follow-up |
| | | visit. No additional lenses will be |
| | | dispensed. |
| | · | A new lens will be opened and worn |
| | | each day. |
| | | Instruct the subject to bring back all |
| | | Unworn study lenses |
| | | Instruct the subject no cleaning or |
| | | disinfecting solutions will be used. If |
| | | determined necessary by the |
| | | Investigator sterile non-preserved |
| | | rewetting drops may be dispensed to |
| | | be used as needed for dryness. |
| | | Subjects will be instructed to wear |
| | | lenses for a minimum of 6 hours a day, |
| | | every day during the study. |
| | | Subjects will be instructed to wear their classes when not wearing the |
| | | their glasses when not wearing the |
| | | study lenses. |
| | | Note: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly |
|---|---|---|
| 2.19. | Schedule Follow-up<br>Visit | differentiated from the other worn lenses that will be shipped back to the Sponsor. The subject will be scheduled to return for their follow-up appointment in 7±1 days. Instruct the subject to bring their habitual contact lenses or glasses to Visit 3. No lenses will be dispensed at Visit 3. |

# VISIT 3

The subjects must present to Visit 3 wearing the study lenses.

| | Visit 3: Treatment 1 Follow-Up 2 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 3.1 | Adverse Events, | Review the subject's concomitant medications | |
| | Medical History and | and record any changes from the previous | |
| | Concomitant | study visit. | |
| | Medications Review | Record any adverse events or medical history | |
| | | changes from the previous study visit. | |
| 3.2 | Wearing Time | Record the average wearing time and | |
| | | comfortable wearing time. | |
| 3.3 | Compliance | Confirm compliance with the prescribed wear | |
| | · | schedule. | |
| ] | | Note: Subjects must have worn lenses for at | |
| | | least 6 hours per day. | |
| | | To be counted as a day of wear at this visit the | |
| | | Subject must have worn the study lenses for 6 | |
| | | hours prior to the visit. | |
| 3.4 | PRO and CLDEQ-8 | The subject will evaluate the vision | |
| | Questionnaires | characteristics, comfort characteristics, | |
| | | handling characteristics, and visual symptoms | |
| | | of the study lenses using the PRO | |
| | | questionnaire and the Contact Lens Dry Eye | |
| | | Questionnaire | |
| 3.5 | Subject Reported | Subjects will respond to a verbal open-ended | |
| | Ocular Symptoms | symptoms questionnaire. | · |

| 3.6 | Visual | Record whether the subjects distance and near | |
|---|---|---|---|
| 3.7 | Satisfaction Distance and Near Entrance Visual Acuity | vision with the lenses is acceptable. Measure the distance and near visual acuity OD, OS and OU to the nearest letter. Record the results. | |
| | | Note: Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity | |
| 3.8 | Binocular Over-<br>refraction | Perform a binocular over-refraction and record<br>the OD and OS results and distance visual<br>acuity. | Appendix<br>F |
| | | Note: No lens changes are allowed based on the over-refraction. | |
| 3.9 | Lens Fit<br>Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). • The subject should not proceed to wear the lenses if any of the following is observed: | |
| | | <ul> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> </ul> | |
| | | <ul> <li>presence of unacceptable movement<br/>(excessive or insufficient) in all three<br/>movement categories (primary gaze,<br/>upgaze, and push-up).</li> </ul> | |
| | | If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. | |
| 3.10 | Visual Performance | Visual performance will be recorded OD, OS and OU for the following: Distance, Bright Illuminance ETDRS Charts 3M-HC#1, HC#2, HC#3 and LC#1, LC#2 and LC#3 | |
| | | Near, Bright Illuminance<br>Reduced Guillon-Poling charts<br>High Contrast and Low Contrast Intermediate<br>(64cm) and Near (40cm). | |

| | 1 | Distance Dim Illuminance | |
|---|---|---|---|
| | | Distance, Dim Illuminance | |
| | | (with Distance goggles) | , |
| | | ETDRS Charts 3M-HC#4, HC#5, HC#6 | |
| | | Near, Dim Illuminance | |
| | | (with Near goggles) | |
| | | Reduced Guillon-Poling charts | |
| | | High Contrast | |
| | | Intermediate (64 cm) and Near (40 cm). | |
| | | intermediate (or only and real (re only). | |
| | | Note: | ı |
| | | The room illuminance must be between | |
| | | 7.3 and 7.9 EV. | |
| | | Distance, HC-1 Chart luminance | |
| | | Acceptable EV Range 10.5-10.7. | |
| | | Guillon-Poling, Near Chart luminance | |
| | | Acceptable EV Range 10.8-11.1. | |
| | | Do not use the Mesopic filter for Dim | |
| , | • | luminance (Dim luminance will be | |
| | | simulated by using the goggles) | |
| 3.11 | Collection of | Collect unworn lenses returned by the subject. | |
| 3.11 | unworn lenses | Confect unworm renses returned by the subject. | |
| 2.12 | Lens Removal | The study lenses can be removed, and saved in | |
| 3.12 | Lens Removai | sterile saline in labeled glass vials | |
| 2.12 | Diaminana | FDA Slit Lamp Classification Scale will be | |
| 3.13 | Biomicroscopy | • | |
| | | used to grade the findings and determine | |
| | | eligibility. For the conjunctival redness 0.5 | |
| <b>.</b> | | 1 02 422 5523 4225 5 | |
| | | unit increments will be used in the grading. | |
| | | Corneal Staining Assessment will | |
| | | be graded in 1.0 increments. | i |
| : | | If the clearance of the fluorescein needs to be | |
| | | expedited, preservative-free rewetting drops or | 1 |
| 1 | | saline may be instilled. | |
| 3.14 | Exit Distance and | Distance and near Snellen visual acuity will be | |
| | Near Visual Acuity | measured for each eye with the subject's | |
| | | habitual correction in place. | |
| | | * | |
| | | For near measures use the ETDRS 2000 Series | |
| | | Chart 1 or 2. The acuity will be recorded to the | |
| | | nearest letter OD, OS and OU. | |
| 3.15 | Wash-out | Subject will complete a 6±2 days wash-out | |
| 3.13 | Period | period during which they can wear their | |
| | 1 Citod | habitual contact lenses or glasses. | |
| 1 | | madition comment formers of Emphosis | I |

| Note: Instruct the Subject to report to Visit 4 |
|-------------------------------------------------|
| wearing their habitual contact lenses. |

Visit 4
Subjects must report to this visit wearing their habitual contact lenses, to accurately assess baseline CLUE performance. If the subject is not wearing their lenses they must be rescheduled.

| resched | Visit 4: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 4.1 | Adverse Events, Medical History and Concomitant Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. |
| 4.2 | Baseline Questionnaire and CLDEQ-8 Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of their habitual lenses using the PRO questions and the Contact Lens Dry Eye Questionnaire |
| 4.3 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 4.4 | Entrance Distance<br>and Near Visual<br>Acuity | Record the distance and near Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual contact lens correction in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 4.5 | Lens Removal | Have the subject remove their habitual lenses and store in an approved solution. |
| 4.6 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. For the conjunctival redness (1) 0.5 unit increments will be used in the grading. Corneal Staining Assessment (1) will be graded in 1.0 increments. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 4.7 | Continuance | Determine whether the subject is eligible to continue in the study based on the examination findings. |

| | | Visit 4: Treatment 2 Lens Fitting | |
|---|---|---|---|
| Step | Procedure | Details | |
| 4.8 | Lens Selection | Select the lens pair and power based on the randomization table and appropriate fitting guide for each eye. Record the test lens parameters (power and lot number). | Appendix G or H Fitting Guides |
| 4.9 | Lens Insertion | The Investigator or the subject inserts the study lenses. Record the time of lens insertion. Check for lens damage under the slit lamp before proceeding with lens settling. Replace damaged lenses if applicable. Worn, damaged lenses must be saved in saline and a product complaint form completed. | |
| 4.10 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. | |
| 4.11 | Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. | |
| 4.12 | Distance and Near<br>Visual Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. Note: Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity | |
| 4.13 | Over-refraction | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 4.14 | Lens Fit<br>Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The subject will not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze | |

| | | | - |
|---|---|---|---|
| | | <ul> <li>presence of edge lift</li> <li>presence of unacceptable movement<br/>(excessive or insufficient) in all three<br/>movement categories (primary gaze,<br/>upgaze, and push-up).</li> </ul> | |
| ļ | | If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation | |
| 4.15 | Modifications | If the subjects vision is unacceptable for at least one distance or the Investigator determines that the visual acuity or overrefraction are not acceptable then a lens modification must be made. Up to two attempts at modification are permitted if necessary, to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the appropriate fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. If modifications are required steps 4.8 to 4.14 will be repeated for each modification. | Appendix G or H Fitting Guides |
| 4.16 | PRO Post-Fit<br>Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of their study lenses using the PRO questionnaire. | |
| 4.17 | Exit Distance and<br>Near Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. Note: The distance visual acuity must be at | |
| 4.18 | Dispensing<br>Criteria | <ul> <li>least 20/30 OU for the lenses to be dispensed.</li> <li>The lenses will be dispensed for 2-4 days.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> </ul> | |

| | | Subject must indicate that the comfort |
|---|---|---|
| | | of the lenses is acceptable. |
| | | Lenses must have an acceptable |
| | | general lens fit. |
| 4.19 | Subject | Instruct the Subject the following: |
| | Instructions | The lenses will be worn on a daily |
| | | wear basis. |
| | | Only enough lenses will be dispensed |
| | | to the subject to wear for the required |
| | | number of days until their follow-up |
| | | visit. No additional lenses will be |
| | | dispensed. |
| | | A new lens will be opened and worn each day. |
| | | <ul> <li>Instruct the subject to bring back all</li> </ul> |
| | | Unworn study lenses |
| | | Instruct the subject no cleaning or |
| | | disinfecting solutions will be used. If |
| | | determined necessary by the |
| | | Investigator sterile non-preserved |
| | | rewetting drops may be dispensed to be |
| | | used as needed for dryness. |
| | | Subjects will be instructed to wear |
| | | lenses for a minimum of 6 hours a day, |
| | | every day during the study. |
| | | Subjects will be instructed to wear their glasses when not wearing the study. |
| | | glasses when not wearing the study lenses. |
| | | icrises. |
| | | Note: In the event a lens is lost or damaged, |
| | | the subject will return to the clinical site for |
| | | replacement. As much as reasonably possible, |
| | | a damaged lens and packaging should be |
| | - | returned to the clinical site (wet, if possible) |
| | | and then returned to the Sponsor. If lens |
| | | damage is present, complete the Product |
| | | Quality Complaint Form. The lens will be |
| | | stored in labeled vial with saline, and clearly |
| | | differentiated from the other worn lenses that |
| 4.20 | Schedule Follow- | will be shipped back to the Sponsor. The subject will be scheduled to return for |
| 1.20 | up Visit | their follow-up appointment in 3±1 days. |
| | | and the specific in the state of the specific in the specific |
| | | Note: To count the follow-up visit as a day of |

| wear the Subject must have worn the study |
|-------------------------------------------|
| lenses for 6 hours prior to the visit. |

# VISIT 5

The subjects must present to Visit 5 wearing the study lenses.

| | | Visit 5: Treatment 2 Follow-Up 1 |
|---|---|---|
| Step | Procedure | Details |
| 5.1 | Adverse Events, | Review the subject's concomitant medications |
| | Medical History and | and record any changes from the previous |
| | Concomitant | study visit. |
| | Medications Review | Record any adverse events or medical history |
| | | changes from the previous study visit. |
| 5.2 | Wearing Time | Record the average wearing time and |
| | | comfortable wearing time. |
| 5.3 | Compliance | Confirm compliance with the prescribed wear |
| | 1 | schedule. |
| | • | |
| | | Note: Subjects must have worn lenses for at |
| | | least 6 hours per day. |
| | | To be counted as a day of wear at this visit the |
| | | Subject must have worn the study lenses for 6 |
| | | hours prior to the visit. |
| 5.4 | PRO and CLDEQ-8 | The subject will evaluate the vision |
| | Questionnaires | characteristics, comfort characteristics, |
| | | handling characteristics, and visual symptoms |
| | | of the study lenses using the PRO |
| | | questionnaire and the Contact Lens Dry Eye |
| | | Questionnaire |
| 5.5 | Subject Reported | Subjects will respond to a verbal open-ended |
| 2.5 | Ocular Symptoms | symptoms questionnaire. |
| 5.6 | Visual | Record whether the subjects distance and near |
| 6.7 | Satisfaction | vision with the lenses is acceptable. |
| 5.7 | Distance and Near | Measure the distance and near visual acuity |
| | Entrance Visual | OD, OS and OU to the nearest letter with the |
| | Acuity | study lenses in place. Record the results. |
| | | Note: Use the ETDRS 2000 Series Chart 1 or |
| | | 2 near card placed at 40 cm to measure the |
| | | Near visual acuity |
| 5.8 | Distance Over- | Perform a distance over-refraction OD and OS |
| J.0 | refraction and | using loose lenses outside of the phoropter |
| | Distance Visual | under ambient room illumination. The |
| | Acuity | distance over-refraction may also be refined |
| | | under binocular conditions. Record the |
| | | results and distance visual acuity OD and OS. |
| l | I | 1 und distutive riduit worthy of stille oo. |

| | | The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
|---|---|---|---|
| 5.9 | Determination of Lens Optimization | If the subjects vision is unacceptable for at least one distance or the Investigator determines that the visual acuity or overrefraction are not acceptable then a lens modification must be made. Up to two attempts at modification are permitted if necessary, to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the appropriate fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. | Appendix<br>G or H<br>Fitting<br>Guides |
| 5.10 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). • The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. | |
| 5.11 | Collection of unworn lenses | Collect unworn lenses returned by the subject when lens power has been optimized. Note: If lens power was not changed allow the subject to use the unworn lenses dispensed at Visit 4 and dispense enough lenses of the same power to last the subject until their next visit. | |
| 5.12 | Lens Removal | The optimized study lenses will be removed and discarded. | |

| C 10 | D: : | TED A CILLY CILLOS IS C. 1 1111 |
|---|---|---|
| 5.13 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. For the conjunctival redness 0.5 unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 5.14 | Insertion of Study<br>Lenses | Dispense the subject new lenses that match the Distance and ADD power of the lenses that were removed in Step 5.12 above. Dispense enough lenses to last the subject until their next visit. |
| 5.15 | PRO Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of their study lenses using the PRO questionnaire. |
| 5.16 | Exit Distance and<br>Near Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 5.17 | Dispensing<br>Criteria | <ul> <li>The lenses will be dispensed for 6-8 days.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> |
| 5.18 | Subject<br>Instructions | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> </ul> |

| | | <ul> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all Unworn study lenses</li> <li>Instruct the subject no cleaning or disinfecting solutions will be used. If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> </ul> |
|---|---|---|
| | | Note: In the event a lens is lost or damaged, the subject will return to the clinical site for replacement. As much as reasonably possible, a damaged lens and packaging should be returned to the clinical site (wet, if possible) and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. |
| 5.19 | Schedule Follow-up<br>Visit | The subject will be scheduled to return for their follow-up appointment in 7±1 days. |

# VISIT 6

The subjects must present to Visit 6 wearing the study lenses.

| | Visit 6: Treatment 2 Follow-Up 2 | |
|---|---|---|
| Step | Procedure | Details |
| 6.1 | Adverse Events, Medical History and Concomitant Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 6.2 | Wearing Time | Record the average wearing time and comfortable wearing time. |
| 6.3 | Compliance | Confirm compliance with the prescribed wear schedule. |

JJVC CONFIDENTIAL

| | | Note: Subjects must have worn lenses for at least 6 hours per day. To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 | |
|---|---|---|---|
| | | hours prior to the visit. | |
| 6.4 | PRO and CLDEQ-8<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire and the Contact Lens Dry Eye Questionnaire | |
| 6.5 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 6.6 | Visual<br>Satisfaction | Record whether the subjects distance and near vision with the lenses is acceptable. | |
| 6.7 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU to the nearest letter. Record the results. | |
| | | Note: Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity | |
| 6.8 | Binocular Over-<br>refraction | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. | Appendix F |
| | | Note: No lens changes are allowed based on the over-refraction. | |
| 6.9 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). • The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). | |
| | | If either lens is deemed unacceptable, the subject will be discontinued from the study. | |

| | | Remove the lenses, perform a slit-lamp | |
|---|---|---|---|
| | | evaluation, and complete the Final Evaluation | |
| | | 1 | |
| 6.10 | Visual Performance | form. Visual performance will be recorded OD, OS | |
| 0.10 | Visual Performance | and OU for the following: | |
| | | Distance, Bright Illuminance | |
| | | ETDRS Charts 3M-HC#1, HC#2, HC#3 and | |
| | | LC#1, LC#2 and LC#3 | |
| | | Near, Bright Illuminance | |
| | | Reduced Guillon-Poling charts | |
| | | High Contrast and Low Contrast Intermediate | |
| | | (64cm) and Near (40cm). | |
| | | (O-TOTI) and I Total (Total). | |
| | | Distance, Dim Illuminance | |
| | | (with Distance goggles) | |
| | | ETDRS Charts 3M-HC#4, HC#5, HC#6 | |
| | | , , | |
| | | Near, Dim Illuminance | |
| | | (with Near goggles) | |
| | · | Reduced Guillon-Poling charts | |
| 1 | | High Contrast | |
| | | Intermediate (64 cm) and Near (40 cm). | |
| | | Note: | |
| | | The room illuminance must be between | |
| | | 7.3 and 7.9 EV. | |
| | | Distance, HC-1 Chart luminance | |
| | | Acceptable EV Range 10.5-10.7. | |
| | | Guillon-Poling, Near Chart luminance | |
| | | Acceptable EV Range 10.8-11.1. | |
| | | Do not use the Mesopic filter for Dim | |
| | | luminance (Dim luminance will be | |
| | | simulated by using the goggles) | |
| 6.11 | Collection of | Collect unworn lenses returned by the subject. | |
| | unworn lenses | | |
| 6.12 | Lens Removal | The study lenses can be removed, and saved in | |
| | | sterile saline in labeled glass vials | <u> </u> |
| 6.13 | Biomicroscopy | FDA Slit Lamp Classification Scale will be | |
| | | used to grade the findings and determine | |
| | | eligibility. | |
| | | For the conjunctival redness 0.5 | |
| | | unit increments will be used in the grading. | |
| | | Corneal Staining Assessment will | |
| | | be graded in 1.0 increments. | |

| If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or |
|---|
| saline may be instilled. |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

Note: If the subject is a screen-failure and a refraction and/or biomicroscopy procedure has just been performed, you may intentionally blank out these forms at the Final Evaluation in EDC.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Subjective<br>spherocylindrical<br>Refraction | Perform subjective spherocylindrical refraction with a phoropter and record the best corrected distance visual acuity to the nearest letter (OD, OS, OU). |
| F.2 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study indicate the reason. |

## 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| Step | Procedure | Details |
|---|---|---|
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit |
| U.2 | Change of Medical History and Concomitant Medications | Questions regarding the change of subjects' medical history and concomitant medications. |
| U.3 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| U.4 | Entrance VA | Record the entrance distance and near visual acuity (OD, OS and OU) to the nearest letter. |
| U.5 | Subjective Sphero-<br>cylindrical<br>Refraction | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. Record the refraction and distance visual acuity to the nearest letter. |
| U.6 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. For the conjunctival redness 0.5 unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| U.7 | Lens Dispensing | Additional lenses may be dispensed if the subject loses, tears, or runs out of lenses. |
| U.8 | Exit Visual Acuity | Record the subject's exit distance and near visual acuity (OD, OS and OU) to the nearest letter. |

# 7.4. Laboratory Procedures

Not Applicable

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

## 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent;
- they are eligible;
- have not withdrawn/discontinued for any reason described in Section 8.2;
- Complete all study visits

## 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to protocol
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2
- Collect all unused test article(s) from the subject

An additional subject may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

## 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications for this study include: Any ocular medications except for rewetting drops.

Concomitant therapies that are disallowed include: Any therapies that may contraindicate lens wear.

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

#### 11. STUDY TERMINATION

If more than 2 subjects in the investigational soft contact lens group develop serious expected (e.g., definite or probable MK) or unexpected device related adverse events, the study will be suspended. Upon review and consultation with IRB, and JJVC safety review committee, the study may be terminated.

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

## 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)".
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or subject)
- OD/OS indication, along with whether or not the lens was inserted
- Any related AE number if applicable

- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eye Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return (

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

Adverse Event (AE) – An AE is any untoward (unwanted) medical occurrence in a patient or clinical investigation subject administered a test article, study treatment or study procedure whether caused by the test article, study treatment or procedure. An AE can therefore be any unfavorable or unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of the test article, study treatment, or study procedure whether or not related to the test article, study treatment, or study procedure.

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study
- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

Serious Adverse Event (SAE) – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the subject's body)
- Is a congenital anomaly/birth defect, or

Requires intervention to prevent permanent damage (the use of the test article resulting in a condition which requires medical or surgical intervention to preclude permanent impairment of the body structure or a body function). Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of >2 Lines of BSCVA
- Other Grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation >2 weeks

**Non-Significant Adverse Events** – Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

Adverse Device Effect (ADE) – A sub-set of AEs, and include only those adverse events that are cause by or related to the investigational device.

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

#### 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; doubtful; possible; probable; very likely see definition in Section 13.2.1)
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events see definition in Section 13.2.2).
- Outcome Not Recovered or Not Resolved; Recovering or Resolving; Recovered or Resolved with Sequelae; Recovered or Resolved; Death Related to Adverse Event; Unknown
- Actions Taken None; temporarily discontinued; permanently discontinued; other action taken

#### 13.2.1 Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article, study treatment, or study procedure. The test article, study treatment or study procedure relationship for each adverse event shall be determined by the Investigator using these explanations:

• Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.

- Doubtful An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is unlikely.
- Possible An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Probable An adverse event that might be due to the use of the test article. The relationship in time is suggestive (e.g. confirmed by de-challenge). An alternative explanation is less likely, e.g. concomitant treatment or concomitant disease(s).
- Very Likely An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

## 13.2.2 Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities

## 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom)
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset
- Date and time of resolution
- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)
- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment /eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether or not a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event /eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator.

## 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event.


In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether or not the adverse event was considered to be related to the test article, study treatment or study procedures.

## 13.4.1 Reporting Adverse Events to Sponsor

## Serious/Significant Adverse Events

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

## Unanticipated (Serious) Adverse Device Effect (UADE)

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

#### 13.4.2 Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set


forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

#### 13.5. Event of Special Interest

None

#### 13.6. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

## 14. STATISTICAL METHODS

#### 14.1. General Considerations

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (Descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation (SD), median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

Summaries will be presented by study lens type and will be performed separately by completion status. All analyses will be conducted on per-protocol population (see section 14.3).

#### 14.2. Sample Size Justification

A total of approximately 80 eligible subjects will be enrolled into the study at this site and at least 60 subjects will complete this study. This is a pilot study for assessing the test articles. As such, the sample size calculation was not based on any power analysis with regard to the primary endpoint. The collected data will be used to design future trials.


#### 14.3. Analysis Populations

# **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

## **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the per-protocol population set will be documented in a memo to file.

## **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

## 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%. No adjustment for multiple comparisons will be conducted unless specified otherwise. This is a pilot study and all the hypotheses are exploratory in nature.

## 14.5. Primary Analysis

Primary efficacy analysis:

## Visual Performance:

Near and distance binocular, high luminance, high contrast visual performance on logMAR scale will be analyzed separately using a linear mixed model to test for the difference between the study lens systems. Each model will include the experimental design factors: sequence of lens wear, lens wearing period and lens type as fixed effects. Other baseline characteristics known of importance such as age, gender, and/or add power will be included as fixed covariates when appropriate. The covariance between residual errors from the same subject across lens wearing periods will be selected based on the finite-sample corrected Akaike's Information Criterion (Keselman et al. 1998). Covariance structures considered may include: Homogenous compound symmetry (CS) and Unstructured covariance structure (UN). The structure that returns the lowest Akaike Information Criteria Corrected (AICC) will be selected as the structure that best fit the data.

Comparisons will be carried out using 95% confidence intervals constructed of least squared means (LSM) from the linear mixed models. Statistical superiority will be concluded if the upper limit of the confidence intervals of the test lens is below +0.01 logMAR for distance and +0.17 for near.


## 14.6. Secondary Analysis

#### **CLUE Vision Score:**

Overall quality of vision scores will be analyzed using a linear mixed model adjusting for baseline values as fixed covariates. The model will include the experimental design factors: sequence of lens wear, period, lens type as fixed effects. The covariance between residual errors from the same subject across lens wearing periods will be selected based on the finite-sample corrected Akaike's Information Criterion (Keselman et al. 1998). Covariance structures considered may include: Homogenous compound symmetry (CS) and Unstructured covariance structure (UN). The structure that returns the lowest Akaike Information Criteria Corrected (AICC) will be selected as the structure that best fit the data.

Comparisons will be carried out using 95% confidence intervals constructed of least squared means (LSM) from the linear mixed models. Statistical superiority will be concluded if the lower limit of the confidence intervals of the test lens is above 32 points.

In all models, the Kenward and Roger method (Kenward and Roger, 1997) will be used for the calculation of the denominator of degrees of freedom.

### 14.7. Other Exploratory Analyses

Not applicable.

#### 14.8. Interim Analysis

Not Applicable

## 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 5 imputations.

# 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

## 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

# 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an Bioclinica Express version 5.5 EDC system. An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

External Date Sources for this study include: Not Applicable

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.

#### 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 16. DATA MANAGEMENT

## 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

# 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study about the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

#### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for monitoring and auditing by JJVC and for inspection by local and regulatory authorities.


#### 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies
- Clarifying questions regarding the study
- Resolving study issues or problems that may arise
- Reviewing of study records and source documentation verification in accordance with the monitoring plan

## 18. ETHICAL AND REGULATORY ASPECTS

#### 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

#### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP), and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013 and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP), and applicable regulatory requirements.


# 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved subject recruitment materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol amendments that increase subject risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki, current ICH and GCP guidelines, applicable regulatory requirements, and Sponsor policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

#### 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Data Protection Act of 1998 and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations. The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential

## 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines, the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP Section 8, Essential Documents for the Conduct of a Clinical Trial, and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will

accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

## 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Investigator's Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

Case Report Forms will be completed in real time according to the study procedures specified in the study protocol. Case Report Forms should be completed and reviewed and signed as applicable by the Investigator within 3 days of visit completion. Data queries must be addressed with complete responses within 3 days of generation. JJVC reserves the right to withhold remuneration until these activities are addressed.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study
- Scheduling a study visit outside the subject's acceptable visit range

#### 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor

## 22. REFERENCES

1. Keselman HJ, Algina J, Kowalchuk RK, Wolfinger RD. A Comparison of Two Approaches for Selecting Covariance Structures in the Analysis of Repeated Measures. *Communications in Statistics—Simulation and Computation*. 1998;(27):591–604.

# APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)












Protocol 5860









































30







Confidential



## APPENDIX B: PATIENT INSTRUCTION GUIDE

Provided separately.
### APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

# PACKAGE INSERT / FITTING GUIDE

### BAUSCH-LOMB

BAUSCH-LOMB

(nesofficon A)
Soft (Hydrophilic)
Contact Lenses ONEday

ONEday or Feed South (nesofficon A) Soft (Hydrophilic) Contact Lenses

RONLY

BAUSCH ...

CAUTION: Foderal law restricts this device to sale by or on the order of a licensed practitioner.

© Baxch & Lomb incorporated.
All dights reserved worldwide.

© ITM are trademarks of
Bastch & Lomb incorporated
or its affiliates. Any other product/
and names are trademarks of
likeir respective owners.

Name and Address of Manufacturer: Beusch & Lomb Incorporated HOO North Geodinan Street Rochester, New York, USA 14609

ONEday (nesofficon A) Soft (Hydrophilic) Contact Lenses

Printed in the U.S.A.





Long term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as servicemental conditions faitured, geography, dout over 3 and personal factors (extent and nature of cuttoors activities). UV blocking contact lenses help provide protection against harmfall UV residence.

\$ S

Warning

UV absorbing contact lenses are NOT substitutes for protective UV absorbing
eyevers untuals. VV absorbing googles or simplesses because they do not
completely cover the eye and surrounding area. You should continue to Lee UV
absorbing eyevear as directed.

The effectiveness of wearing UV absorbing contact lerses in preventing or reducing the inclusions of could disorders associated with exposure to UV light has not been before additional statements associated with exposure to the proper of the count of the waring UV blocking contact lerse is reduce he risk of developing catarats or other eye disorders. Consultyour Eye Care Professional for more information other eye disorders.

The Molical transmittance profile of nessofficon Å lenses vs a Human Cornea and -tuman Lens:

Nesofilcon A Lens -Nominal Center Thickness Offmm (-1.25D)

Cornea—Human Cornea from a 24-year-old person as described in Lerman, S., Radiant Energy and the Eye, MacMillan, New York, 1980, p.58, fig. 2-21.

Lens-Human crystaline lens from a 25-year-old person as described in Waxier M., Fitchins V.M., Optical Radiation and Visual Health, CRC Press, Boca Raton, Florida, 1986, p. 19, fig. 5.

# SYMBOL REFERENCE GUIDE For label and carbons.

| Fee Paid for Waste<br>Management | De In Date | (Expiration Date) | Batch Code | Diameter | Diopter<br>(Lens Power) | BaseCurve | Low or High<br>Add Power | Sphere Power<br>(Diopters) | Cylinder Axis<br>(Degrees) | Cylinder Power<br>(Diopters) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| € | ) i | EXP(EX) | Þ | DIA Ø <sub>T</sub> | PWR (F'v) | BC | ADD | SPH | ΑX | CYL | |
| Do Not Reuse | Temperature<br>Limitation | Shadle Using | Steam or Dry Heat | See Instruction<br>Leaflet | Indicates the | Marking and the<br>Notified Body | Number<br>Authorized | Representative<br>in European<br>Community | Caution: Federal<br>law restricts this | device to sale by<br>or on the order<br>of a licensed | practitioner |
| <b>⊗</b> | 4 | • | SIEHILE ! | $\triangleleft$ | C € 0050 | | | EC REP | R ONLY | | |

| ure<br>ure | | |
|---|---|---|
| | EXP(2) | Use by Date<br>(Expiration Date) |
| ing<br>Dry Heat | LOT | Batch Code |
| nction | DIA Ø <sub>T</sub> | Diameter |
| e l | PWR (F'v) | Okopter<br>(Lens Power) |
| and the<br>lock | ရှင | Base Curve |
| 70 | ADD | Low or High<br>Add Power |
| tative<br>ity | SPH | Sphere Power<br>(Diopters) |
| ederal<br>ts this | ΑX | Cylinder Axis<br>(Degmes) |
| sale by<br>order<br>ed | CVL | Cylinder Power<br>(Diopters) |
| | YYYYMMDD | Effective Date |



# LENS PARAMETERS AVAILABLE The Bausch + Lomb Biotrus = ONEday (presedition A) Soft (14 drophilic) Contact Lers is a homispherical shell of the following dimensions:

| Danneter: Center Thickness: Base Curve: Powers (Sphorical): Powers (Prestly opia) | M.2mm<br>A.5mm (Asignastan)<br>O.65mm to 0.75mm (varies with power)<br>B.5mm<br>B.4mm (Asignastism)<br>G.6001to-6,0001a (0.650) seps<br>-6,5001to-9,0001a (0.650) seps<br>-6,0001to-9,0001a (0.650) seps |
|---|---|
| Add Powers: Powers (Astigmadsm): Cylinder Powers: Auis Additional parameters may t | Add Powers Low (402/Dibt o-1500) and Hgh (4175Dn o-2500) Powers (Astignation): -4.000 to-6.000 in 0.250 taso; Cylleder Powens: Que 1802 Additional parameters may be introduced own time, check for product availability. |

## ABLE OF CONTENTS

scription

MPORTANI

| Lens Parameters Available | ın |
|-------------------------------------------------------|---------------|
| How the Lans Works (Actions) | ø |
| | 40 |
| Crotesingle-shows (Resone Notto) Ital | |
| XXX (HTX) | • |
| Thecautions | œ |
| Adverse Reactions | É |
| Important I setment Information for Adverse Reactions | ; <b>3</b> == |
| | Ŋ |
| Fitting Procedure | £ |
| Pre-Fitting Examination | α |
| Initial Lens Power Selection | Œ |
| Initial Lens Evaluation | Œ |
| Criteria of a Well-Fitted Lens | ന |
| Characteristics of a Tight (Steep) Lens | ¥ |
| Characteristics of a Loose (Flat) Lens | <b>#</b> |
| | ** |
| Practitioner Fitting Sets | ۴Ü |
| | fc. |
| Monoviston Fitting Guidelines | 1 <u>7</u> 2 |
| Select | عوا |
| TVe Selection | 4 |
| Special Fifting Considerations | <b>.</b> |
| dd Detern | æ |
| first Lens Fitting | Φ |
| Adaptation | Q |
| Other Suggestions | 0 |
| Milk Focal Patrice Cuidalines | 2 |
| Parient Selection | 0.0 |
| | 3.5 |
| 4:11 | 3:5 |
| Symptom Resolution | |
| Patient Education | 15 |
| Handing of Lenses | į |
| Sticking (Nonmoving) Lens | 8 |
| | 8 |
| dverse Reactions | 8 |
| How Supplied | 23 |

The Bausch + Lomb Brotne ® ONEday lens material, Hypergus <sup>In</sup> (needizon A), is a hydropinic copolyme of Pythrogweght Inethacytes and Musing providence and sty Staveter by weight when innered in a steel as sime solution. A beroutizone UV. absorbing monomer is incorporated into the manifectuling process to Brotn VV radiation. The transmistrate of the calculation are less than 15% in the UVB range of 250 min of 35cm and less than 50 kin the UVA range of 35cm to 35cm to 35cm to 35cm to 280 min this less is timed blue with Reactive Blue Dyo 246.

The physical / optical properties of the lens are:

8 1374 42x10 "[cm²O<sub>2</sub>(SIP)x cm]/ (secx cm² x mmHg) @ 35° C (Poterographic Method)

Oxygen Permeability (Dk.)

CLE Y value - approximately 99%

Light Transmittance: Spedile Gravity: Retractive Index: WaterContent: The lens is to be prescribed for single-use disposable wear, and is to be discorded after each removal.

should be made available to patients upon request. The eye care professional should provide the patient with the patient instructions that pertain to the patient's prescribed lens and the recommended wearing schedule

DESCRIPTION

This package insert and fitting guide is imended for the eye care professional, but

This package insert and tithing guide has been developed to provide practitioner with information covering describe the ReBasch+ Lonnib Biotrus\*
ONEday (secolifican A) Soft (Hydropthii) Contact lans, Basich + Lonnib Bortus\*
Software Notificative the Percyolasi (encedions) A) Soft (Hydrophiilio) Contact Lans and Basich + Lonnib Biotrus\* ONEday for Assichative A) Soft (Hydrophiilio) Contact Lans and to all laster steef strips operated rest it is electric as of Mydrophiilio) Contact Lans and to all laster steef strips operated rest it is electric as of Mydrophiilio) Contact Lans and to all laster steef strips paredeaters. It is electric as of Mydrophiilio Contact Lans and to all laster steef strips paredeaters. It is electric as of described. Please read consisting and beapt this information for tuture use.

### N

# HOW THE LENS WORKS ACTIONS

The transmittance characteristics are less than 5% in the UVB range of  $280 {\rm Am}$  to 315 nm and less than 50% in the UVA range of 316 nm to 380 nm. In its indicated state, the Bausch + Lorin Brotrus<sup>2</sup> ONEday (needshorn A) Sot (Fydrophilic) Cortext Lase, Barsch + Lorin Brotrus<sup>2</sup> ONEday for Prestycysi (resoftom A) Sott (Hydrophilic) Cortext Lars and Bausch + Lorin Brotrus<sup>2</sup> ONEday for Astigmastin (hecoftom A) Sott (Hydrophilic) Cortext Lars, when placed on the corruss, act as a refracting medium to tocus light rays on the retina.

The Bausch + Lonto Biotrows ONEday (rescalioon A) Soft (14) drophilic) Constact laws is indicated the Pack also were correction of referance an enterpol (myopia, hypercopia and subjurnation) in aphalic and/or non-subhiting peasons with non-diseased eyes, estilability assignastism of 200 dischers or less, that does not interfere with visual south. The less may be prescribed in subserial sowers maping from \*20000 bs-20000. NDICATIONS

The Basseth + Lomb Biotrus® ONEday for Prestyopia (nesoffican A) Soft (Flydroppiilo). Contact Lease in indicated for they wear for the correction of refractive ametropia (myonia, typeropsi) and assignation and greetappial in aphalic and/or non-aptivatic persons with non-diseased eyes, enhibiting assignation of 2020 dispets or less that does not literative with visual acutily. The less may be prescribed in power ranging from +2000D to -2000D with add power ranging from +2000D to -2000D with add power ranging from +2000D to -2000D with add power ranging from +2000D to -2000D with add power ranging from +2000D.

The Bausch + Lomb Biotrue® ONEdayfor Astigmation (needloon A) Soft ("Autopullo,") Context less in siciated for daily west for the connection of foreign the indicated for adjuly west for the connection of foreign by previous and assignation is obtained and on advantage are reconstructing from diseased eyes, exhibiting astigmatism of up to 5000 diopers, that does not infestion with visual scale, in hele may be prescribed in powers in aging it on the ADOXD to -QUOXD to diply west.

The lens is to be prescribed for single-use disposablewear, and is to be discarded after each removal.

# CR-5860, v3.0 Amendment 2.0

ĸ

CONTRAINDICATIONS
(REASONS NOT TO USE)
DONOTUSE the Basset, whom's bounder (needlean A) Soft
(Photophia:) Central Lenn's Browne' ONEsty (needlean A) Soft
(Photophia:) Central Len, Basset, who Bistrae CoNEsty for Presbypsia
(reasoften A) Soft (Phytophia:) Central Lens or Basset, when Belorue'
ONEsty for Astyrmatican (needlean A) Soft (Phytophia:) Central Lens when
any of the following conditions estit.

- Acute and subscute inflammation or infection of the anterior chamber of
- Any eye disease, injury, or atmormality that affects the comes, conjunctive, or eyelids

  - Severe insufficiency of lacrimal secretion (dry eyes)
    - Comesi hypoesthesia (reduced corneal sensitivity)
- Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses
- Allergia reactions of ocular surfaces or adnexa (surrounding tissue) that may be influeed or exagged ted by wearing contact lenses or use of contact lens solutions
  - Any active comed infection (bacterial, fungal, or viral)
  - if eyes become red or initated

### WARNINGS

After a thorough eye examination, including appropriate medical background, packens should be tully appreciately the prescribing professional of all the fits with contact leave wen. Externis should be advised of the following warmings perfaining to contact leave wear:

- Problems with contact lense and lens care products could result in serfores injusy to the eye. It is essential that patients follow these eye care prodessionals direction and all albeing instructions for proper use of lense and lens care recoults, including the lens case, they problems, including contreal when can develop neptily and lead to losts of vision.
  - Daily wear lenses are not indicated for overnight wear, and patients thould be instructed forth overal lenses while steeping. Clinical studies have shown that the risk of serious adverse neartiers is increased when daily wear lenses away no vernight.
    - Studies have shown that contact lens wearens who are smokers have a higher incidence of adverse reactions than porsmokers.

- if a patient experiences eye discomfort, excessive tearing, vision changes, or redness of the eye, the patient should be instructed to **insmediately remove lenses** and promptly contact his or her eye care professional.
- Patients should be instructed not to expose their contact lenses towerentiale weering them.
- Water can harbor microorganisms that can lead to serere infaction, vision loss or thingeness if their contact lenses have been submersed in water when sometiming in pools, lakes to contact lenses should be discarded and replaced with a new pair Recommendations for wearing lenses cluring any water activity should be discussed with the patient.

### REGUIONS

# Special Pracavilons for Eya Cara Professionals:

Due to the small number of patients earnibed in clinical investigation of lenses, all enfaction provest, degion configurations, or lens parameters available in the lens makerial are not evaluated in significant numbers. Consouvertly, when electing an appropriate lens design and parameters, the eye care parolessional should excepted and characteristics of the lens that can affect lens parolessional should health, including oxygen permeability, westtability, central and peripheral this canadoptic zone diameter.

- The potential impact of these factors on the patient's cultar health should be carefully weighted against the patients need for which achieves, the confinding oculiar health of the patient and lens per formance on eye should be carefully monitored by the or rescribing eye care professional. Patients who west contact lenses to correct preclycipia may not achieve the best corrected obtained and solutly for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Eve care professionals should instruct the patient to REMOVEA LENS IMMEDIATELY if an eye becomes red or irritated.
- Fluorescein, a yellow dye, should not be used while the lanses are on the ayes. The lanses absorb this dye and become discolored. Whenever fluorescein is used in eyes, the eyes should be flushed with sterile sales solution that is recommended for in-eye use.
  - The patient should be instructed to always discoard disposable larges and larges worn on a frequent/planned replacement schedule after the recommended wearing schedule prescribed by the eye care professional.
- Aswith ary contact letrs, follow-up-visits are necessary to assure the continuing health of the patients eyes. The patient should be instructed as to a recommender follow-up schedule.

- Apri akic parients should not be itted with Bausch + Lomb Biotrue\* ONEday (recardion A) Saft Mydroptials, Combact Hersen, Blanch Lomb Biotrue\* ONEday to Pestyosia-finesolison A) Saft (Mydrophilio) Combact Lerses or Bausch + Lomb Biotrue\* ONEday for Asignasism (nesedion A) Saft (Pydrophilio) Combact Lerses or Bausch + Lomb Biotrue\* ONEday for Asignasism (nesedion A) Saft (Pydrophilio) Contact Lenses until the determination is made that the eye has hasted completely.
- The lenses are prescribed for disposable wear, and are to be disposed of once they are removed from the benefits 49st, littpoor surface placehors be instructed to always have available a paint finesticement lenses. In the event that a lense must be removed from the ege because of dat, a foreign body or other contentinent eyes on the lense of the foreign energy and always and the service and spets on the lense of the foreign energy and always are contentioned and replaced with a replacement lens.

Patients should be advised about wearing lensus during sporting and water related activities. Exposure to water valler wealing contact lensus in activities such as swimming, weder staing and hot then may increase after risk of could militarious including but not times to be deard and the could militarious including but not times to Actarizations be satisfie.

Always contact the eye care professional before using any medicine in the

Never use tweezers or other tools to remove lenses from the lens container unless specifically indicated for that use. Pour the lens into the hand.

As with any contractions, follow-up vists are necessary to assure the continuing health of the eyes. The patient should be instructed as to a recommended follow-up schedule.

Topics to Discuss with the Patient

Who Should Know That the Patient is Wearing Contact Lenses:
Patients should inform their doctor (health care professional) about beings

contact lens wearer.

Patients should always inform their employer of being a contact lers wearen Some jobs may require the use of eye protection equipment or may require that you do not wear lerses.

The patient should be informed that the following problems may occur: Eyes stinging, burning, tiching (tritation), or other eye pain

ADVERSE REACTIONS

Eyecare professionals should carefully instruct posterite about the bollowing safety presentations. It is strongly recommended the posterite be provided with a copy of the Platent Information Bookslation Bases.—Lornho Booture O'Nician (Genezille A) Safeth Vertorial posterior (John Booture O'Nician the Platent Information O'Nician (Larch Booture) (O'Nician to Presty opicial posterior A) Soft (If you opicial careful and Platent I Lenn Borture Wo O'Nician to Do Nician Ford O'Nician to Do Nician Ford A) Soft (If you opicial content Lens and latent from Basesch + Lornho Borture) and understand its contents prior to disponing the lenses.

### Handing Precautions:

- Always weath and rife e hards before handling lentee. Do not get commetics, fortion, season, creams, declorating, or specifie the eye or on the lentee. It is best found on lenses before putting on makeup. Water-base occamefus are less likely to damage lentee than old-base products.
- Be sure that before leaving the eye care professionals office, the patient is able to remove leaves promptly or have someone else available to remove them.

Abnormal feeling of something in the eye (foreign body, scratched area) Excessive watering (tearing) of the eyes

Unusual eye secretions

Redness of the eyes

Blurred vision, rainbows, or halos around objects Reduced sharpness of vision (poor visual acuity)

Sensitivity to light (photophobie)

Comfort is less than when lens was first placed on eye

- Be certain that the fingers or hands are free of foreign materials before touching senses, as microscopic scratches of the lenses may occur, causing distorted vision and/or injury to the eye.
- Always handle lenses carefully and avoid dropping them.
- Do not touch the lens with fingernaits.
- Carefully follow the handling, insertion, removal, dearning distribacting, as storing and weeking instructions in the Planter Harmand bootbeffor the Bausch+Lomb Biotues (Ordicay (nesselincon A) Safe (Hydroptilia) Contral Lerses / Bausch+Lomb Biotues (Ordicay for Presponsis (pescelincon A) Safe (Hydroptilia) Contral Research Lomb Biotues (Ordicay for Astigmatism (insection A) Safe (Hydroptilia) Contral Research Research Lomb Biotues Ordicay for Astigmatism (insection A) Safe (Hydroptilia) Contract Lerses and those prescribed by the system professional.

## 

### 1. Pre-Fitting Examination

 $\mbox{\ensuremath{\ensuremath{\ensuremath}\ensuremath{\ensuremath}\ensuremath{\ensuremath}\ensuremat$ 

The eye care professional should notifit patients who cannot or will not adhere to a recommended one or replacement regimen, or are unable to piece and remove the lenses. Fairer to follow hardling and oleaning instructions could lead to serious eye infectors which might result in corneal ulcors.

Patient communication is vital because it relates not only to patient selection but also to ensure complaince. It is also necessary to discuss the information contained in the Patient information. Booklet with the patient at the time of the initial examination.

• If the discontrion or problem stops, then look closely at the lens. If the lens is in any way dramaged, but not the their back or the sew. These the lens in the storage case and contactine upon expensional. If the lens has diff, an websit, not when their body on the problem notops and the lens appears undampaged, the patient should incoughly clean, fries, and delirled the lenses then retirent them. After retreation, if the problem confirms, the potents should immediately remove the lenses and consult his or har eye care professional.

Here patient notices any of the above, he or she should be instructed to:
Immediately remove the lenses.

- Determine whether a patient is a suitable candidate for contact lenses (consider patient hygiene and mental and physical state),
  - Make ocular measurements for initial contact lens parameter selection, and
- Collect and record baseline clinical information to which post-fitting examination results can be compared.
  - A pre-fitting examination should include spherocylinder refraction and VA, keratometry, and biomicroscopic examination.

Palients selected to wear Bausch + Lomb Biottue® ONE day (neediborn A) Soft (Hydrophiles) Context Lenses, Bausch + Lomb Biottue® ONE day for Prest-boots as Constant Areas or Bausch + Lomb Biottue® ONE day for Astigmatism (needitorn A) Soft (Hydrophile) Context Lenses as should be chosen for their motivation to wear context-lenses, general health and cooperation. By each per care processional most take care in selecting, earmining and eighturching context-lens gaintent. Palent hygiene and willingness to follow gracificorer instructing are essential to their success.

If the above symptoms continue after removal of the lens, or upon reiseardon of a sten, or upon reiseardon of a sten, or upon reiseardon in new float, the lengthest should immediately of a sten, or upon the stendard that the property of the stense and contact his or have see are protesting the more and contact his or have seen protesting the contact his form to enter a stendard the more than the stendard the formation of Adverse Seardons). A serious condition such as infection, controlled they conneal vectors expense and may see the see sections such as a infection, conneal wealth and they conserve a conselve according to the see sections cauch as a brasilon; spellbedist staining or bearership conjunctivity must be managed and treated carefully to avoid more revious

A detailed history is crucial to determining potent needs and expectations. Your patient should be questioned regarding vocation, desired lens vealing time (full or patient), and desired lens usage (reading, recreation or hobbies).

initial evaluation of the utal lens should be preceded by a complete eye examination, including visual acuity with and without correction at both distance and neer, seratomety and sit lenne examination.

- Autial Lans Power Selection
   Lans power is determined from the patient's soherical equivalent prescription corrected to the cornesi plane.
- Select the appropriate here and place on the eye. Aflow the levs to remain on the eye of any age sought (10 to 20 minuse) to achieve a state of equilibrium. Small wartations in the textilety, plf of the less solutions and individual hear composition may cause slight changes in fitting chances risks.
  - Allow ary increase in tear flow to subside before evaluating the ters. The firms required will vary with the individual.
    - 3. Initial Lens Evaluation
- To determine proper lens parameters observe the lens relationship to the eye using a silk lamp.
  - Movement The lens should provide discernible movement with: Primary gaze blink

It is normal for the patient to experience mild symptoms such as lens awareness, variable vision, conscious harm (verlang vers) and slight redenss during the adjustic principal and adjust redenss during the adjustic principal and principal and adjust redensing the adjustic principal article states of though the adjustic principal article states as ymprotrums will disappear.

Important Trustment Information for Advarsa Reactions
Sight-treasening octat complications associated with contactions were can
develop rapidly, and therefore saidy recognition and treatment of proclems
are critical Infectious comes literation is one of the most serious proteins
are critical infectious comes literation in one of the most serious proteins
are critical infections and may be ambiguous in the early tages, States and symptoms of
infectious comes eliceration include discomfort, pair, infarmation, purulent
discharge, sensitivity to light, cells and flare, and comesil infiltrates.

complications

these symptoms persist, the patient should be instructed to contact his or her eye care professional.

Initial symptoms of a minor abrasion and an early infected ulcor are sometimes semilar. Accordingly, usuch spikibile delece, if proteined properly in may develobe, into an intereduction of these conditions, as peter threshold ulcors, in order to revent serious programs on of these conditions as peter threshold ulcors, in order to revent serious programs of the serious programs of the serious programs of the serious order under the serious as potential reduced as perions, the series of serious thresholds as peter paching or the use of steroids or star older inchoice contributions such as expensively or the use of steroids or star older inchoice contributions may examined the error should be entrowed immediately and the ilens and lens care examined the lens and other care products instrined the and entropy in additional star and lens care products instrined to making an order alluthing.

- Upgaze blink
- Centration: The tens should provide full corneal coverage.
- b. Lers evaluation allows the contact lens fitter to evaluate the lens/companies and the same manner as would be done with any soft lens.

### 4. Criteria of a Well-Fitted Lens

if the initial lens selection halfy cowers the cornea, provides discensible movement after a blink is comfortable for the patient and provides satisfactory visual performance, it is a well fitted lens and can be dispensed.

## Characteristics of a light (Steep) Lens

A lean which is much boo steep may subjectively and objectively cause distortion which is much boo steep may subjectively and objectively it seek the rinkal subjective and objective size of the manipular year. But the conflict findings may be quite good. A marginally teep lean may be differentiated from a properly fitted lens by having apprehent pay be differentiated from a properly fitted lens by having apprehent pay to differentiated from a properly fitted lens by having approximately (Dimm while a steep lens will lend to side downward approximately (Dimm while a steep lens will remain relatively stable in relationship to the corneap particularly with the blink.

## 6. Characteristics of a Loose (Flat) Lens

- Decenter, especially on post-blink. if the lens is too flad, it will:
- Have a tendency to edge lift inferiorly and sit on the kower lid, rather than positioning between the sciers and pelipetral conjunctive.
- Have a tendency to be uncomfortable and irritating with fluctuating vision
- Have a tendency to drop or lag greater than  $20 \mathrm{nm}$  on upgaze post-blink.
- Follow-up examinations are necessary to ensure continued successful contact lens wear. From the day of dispensing, the following schedule is a suggested guideline for follow up. Follow-up Care
  - 3-4 days post-dispensing · 10 days
- · 1month
- 3 months
- Every six months thereafter
- At the initial follow-up evaluations the eye care professional should again reassure the patient that any of the previously described adeptive symptoms are normal, and that the adaptation period should be relatively brief.
- Prior to a follow-up examination, the contact lenses should be worn for at least 4 continuous fours and the patient should be asked to blentify any problems which might be occurring related to contact lens wear.
  - With lerses in place on the eyes, evaluate fitting performance to assure that CRITERIA OFA WELL FITTED LENS continue to be satisfied. Examine the lenses dosely for surface deposition and/or damage.

## JJVC CONFIDENTIAL

CR-5860, v3.0 Amendment 2.0

- After the lens removal, instill sodium fluorescein [unless contraindicated] into the eyes and conduct a thorough biomicroscopy examination.
  - The presence of vertical corneal striae in the posterior central comes and/or corneal neovascularization may be indicative of excessive corneal edema.
- The presence of corneal staining and/or limbal-conjunctival hyperemia can be indicative of an unclean lens, a reaction to solution preservatives, excessive lens wear, and/or a poorly fitting lens.
  - 3. Papillary conjunctival changes may be indicative of an unclean and/or damaged lens.

If any of the above observations are judged abnormal various professional judgments are necessary to alleviate the problem and restore the eye to optimal conditions. If the CRITERIA OF A WELL FITTED LENS are not stabilised during any follow-up examination, the patient should be re-fitted with a more appropriate lens.

# PROSE TENONER SERVICES

Lenses must be discarded after single use and must not be used from patient to patient

## WEARING SCHEDULE

There may be a tendency for the daily wear patient to over-wear the lenses initially. Therefore, the importance of addering to a proper, hilled ladywaring schedule should be stressed to these patients. The wearing schedule should be determined by the eye care professional. The wearing schedule chosen by the eye care professional. The waring schedule chosen by the eye care professionals frould be provided to the patient. The lens is to be prescribed for single-t-axe disposable wear, and is to be discarded after each removal. The wearing and replacement schedules should be determined by the eye care professional. Regular checkups, as determined by the eye care professional, are extremely important. Daily Wear

# MONOVISION TITING GUIDELINES

Monovision Needs Assessment for a good part of the state

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual auth) and steeposity) is should be determined by trial whether this patient can function adequately with monovision. Monovision contact lens wear may not be optimal for such activities as:

ند ڼ

Visually demanding situations such as operating potentially dangerous machines yor performing other potentially hazardous activities; and 2. Diving automobilise (e.g., driving at night) Palients who cannot pass their state drivers it carse requirements with monoision correction should be ordived for not drive with this correction. OR may require that additional overcorrection be prescribed.

Visual Demands Method Consider the patients occupation during the eye selection process to determine the critical wison requirements. If a patient's gaze for near tasks is usually in one direction correct the eye on that side for near.

A secretary who places copy to the left side of the desk will usually function best with the near lens on the left eye.

Example:

Special Fitting Considerations

Unidate at Lens Correction

There are circumstances where only one contact lens is required. As an example, an emmercopic patient would only require a near lens while a bilateral myope may

require only a distance lens.

A presbyopic emmetropic patient who requires a +1.75 diopter add would have a +1.75 diopter lens on the near eye and the other eye left without a lens. A presbyopic patient requiring a +150 diopter add who is -2.50 diopters myopic in the right eye and -150 diopters myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.

Patient Education
All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with bitical reading glasses. Each patient should understand that monovision can create a reading glasses. Each patient should understand that monovision can create a reading glasses. Each patient should not extend that monovision can create distance and near tasks. During the fifting process it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision in straight ahead and upward gaze that monovision contact lenses provide. ف

Generally, the non-dominant eye is corrected for near vision. The following test for eye dominance can be used.

a. Ocular Preference Determination Methods

Awass prescribe the lens power for the near eye that provides optimal near acuity at the mitgorin of the patients' habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

4. Near Add Determination

- Method I-Determine which eye is the 'sighting dominant eye.' Have the patient point to an object at the far end of the room. Cover one eye, if the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye.
- Case history and standard clinical evaluation procedure should be used to determine which sets to be corrected for distance and which eye is to be corrected for distance and which eye is to the corrected for near. Next determine the near add. With trial ienses of the proper power in place observe the reaction to this mode. Method 2—Determine which eye will accept the added power with the least reduction in vision. Place a trial spectacle near addlers in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near addlers over the right or left eye. Refractive Error Method For anisometropic corrections, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

A trial fitting is performed in the office to allow the patient to experience monovision correction. Lenses are it according to the directions in the general fitting guidelines.

5. Trial Lens Fitting

Immediately after the correct power lenses are in place, walk across the room and have the patient look at your. Assess the patient reachon to distance vision under these circumstances. Hen have the patient look at lamilar near objects such as a worth deep or fingential, shop and assess the action. As the abelient communes to look around the room at both near and distant objects, observe the reactions. Only after these vision tasks are completed should he patient be asked to read print. Evaluate the patient is eastion to large print (e.g. hyperwritien copy) at first and then graduate to newsprint and finally smaller type sizes. of correction

After the patient's performance under the above conditions are completed, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a guarded prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

Visually demanding situations should be avoided during the initial wearing period. A patient may at this supperences some mild blurred vision, dizziness, headaches, and a feeling of sight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a fried minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process the patient can be advised to first use the lenses in a comfortable familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. In its particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a possenge if its to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

### 7. Other Suggestions

The success of the monovision technique may be further improved by having your patient follow the suggestions below.

- Having a third contact lens (distance power) to use when critical distance viewing is needed.
- Having a third contact lens (near power) to use when critical near viewing is needed.
- Having supplemental spectacles to wear over the monovision contact lenses for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot meet state licensing requirements with a monovision correction.
  - Make use of proper illumination when carrying out visual tasks.
- Success in fitting monovision can be improved by the following suggestions:
- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of the clear near vision in straight ahead and upward gaze with monovision.

CR-5860, v3.0 Amendment 2.0

Q

The decision to fit a patient with a monovision correction is most appropriately left to the eye care professional in conjunction with the patient after carelully considering the patient's needs.

2

All patients should be supplied with a copy of the Bausch + Lomb Biotrus\* ONEday (nesofficen A) Soft (Hydrophilis) Contact Lens. Bausch + Lomb Biotrus\* ONEday for Preshopsi (nesofficen) Soft (Hydrophilis) Contact Lens. Bausch + Lomb Biotrus\* ONEday for Astigmatism (nesofficen A) Soft (Hydrophilis) Contact Lens Patient Information Booklet.

# MULIFOCAL FITING GUDELINES

- Realistic expectations 1. Patient Selection a. Good motivation
  - - 2. Lens Selection
- Determine ocular dominance for distance vision, Update spectacle refraction and Add power.
- Select lens distance prescription based upon spherical equivalent from spectacle prescription, adjusted for vertex distance if necessary. ن
  - Choose trial lenses based upon the above calculation and select Add power. Low Add: +075D to +150D

τi

- High Add: +1,75D to +2,50D
  - 3. Lens Fitting
  - Equilibrate for 10 minutes. ri
- Evaluate distance and near vision binocularly in normal room illumination.
- If vision at distance and near are satisfactory, dispense lenses and schedule follow-up exam within 1-2 weeks.
  - 4. To refine Near Vision
- Refinement 1: Place High Add Iens in non-dominant eye while keeping Low Add Iens in

If patient is wearing two Low Add lenses:

Refinement 2: Hission is still unsatisfactory, continue adding +Q.25D at a time to the non-dominant eye using handheld lenses. Adjust contact lens power when vision in astistactory.

# If patient is wearing two High Add lenses:

4

- Refinement 1: Add +025D to the non-dominant eye.
- Refinement 2:
- If vision is still unsatisfactory, continue adding  $\pm 0.25D$  at a time to the nondominant eye using handheld lenses.

## 5. To refine Distance Vision: If patient is wearing two Low Add lenses:

- Reinnement I: Place SVS lens in dominant eye while keeping Low Add lens in non-dominant
  - Refinement 2:

I vision is still unsatisfactory, add -0.25D at a time to dominant eye using hand held lenses. Adjust contact lens power when vision in satisfactory.

## If patient is wearing two High Add lenses:

- Refinement I:
   Place Low Add lens in dominant eye while keeping High Add lens in non-dominant eye.
- If vision is still unsatisfactory, add -0.25D at a time to dominant eye using hand held lenses. Adjust contact lens power when vision in satisfactory.

### 6. Patient Education

All patients do not function equally well with multifocal correction. Patients may not perform as well for certain tests with this correction as they have with multifocal reading glasses. Each patient should understand that multifocal correction can create a vision compromise that may reduce visual aculty and depth perception for distance and near tasks. During the filting process it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision in straight alread and upward gaze that multifocal contact terses provide.

## HANDLING OF LENSES

### Patient Lens Care Direction

When lenses are dispensed, the patient should be provided with appropriate and advantage instructions and warmings for lens care handling. The eye care professional should recommend appropriate and adequate procedures for each individual patient in accordance with the particular lens wearing schedule.

∞

### CARE FOR A SHICKING (NOMMOVING) LENS

If the lens sticks (stops moving), the patient should be instructed to use a bub-richargo or reweting solution in the feet, the patient should be fasturated to not use plain water, or anything other than the recommended solutions. The patient should be instructed to contact the eye care profession all the text does not begin to move upon binking after several applications on the solution, and to not attempt to remove the lens secogial on the eye care professional.

### 

If Chemicals on wheth Conselector particular case, and an expension paper down of memory obernicals and are spatial of the WATTAND THEN REPROYED FOR PROPERSY PROPINITY TAYNON THE TOWN THEN REPORTSONAL OR VISTA HOSPITAL EMERGENCY ROOM WITHOUT DELAY.

# REPORTING OF AUVERSE REACTIONS

All serious adverse experiences and adverse reactions observed in patients wearing Bander 4- Lornb Bornber (\*O)KEdaylor (\*Red)Roch (\*A)KEdaylor (\*Red)Roch (\*A)KEdaylor (\*Red)Roch (\*A)KEdaylor (\*Red)Roch (\*A)KEdaylor (\*A)KEdayl

Bausch & Lomb Incorporated 400 biomedia Street AdONorth Goodman Street Rochester, New York 14609

Toll Free Telephone Number In the Continental U.S., Alaska, Hawaii 1-800-553-5540

In Canada 1-888 459-5000 (Option 1 - English, Option 2 - French)

### HOW SUPPLIED

Each sterile lens is supplied in a plastic package containing borate buffered saline solution with poloxamine. Each container is marked with the manufacturing lot number of the lens, diopter power, and expiration date.

## JJVC CONFIDENTIAL


ß

8



### DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) Soft

**Contact Lenses for Daily Disposable Wear** 

W900038292

IMPORTANT. This package insert is effective as of March 2016 and applicable to the deleticon A contact lenses described below. Please read carefully and keep this follows:

In this package insert is effective as of March 2016 and applicable to the eye care professional, but should be made available to patients upon nequest. The eye care professional should provide the patient with appropriate instructions that periath to the patient's precribed lenses. Copies of this package insert is available which is recommended to be given to patients.

On the patient instruction Booklet is available which is recommended to be given to patients.

CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed eye care professional.

### PRODUCT DESCRIPTION

DAILIES TOTALI\* and DAILIES TOTALI\* Multifocal (delefficon A) water and 67% (deletilicon A) polymer, a silicone containing hydrogel with added phosphalidytcholine. The core lens material containing 33% water transitions through a water gradient to a hydrogei surface layer that exceeds 80% water. Lenses contain the color additive copper phthalocyanine, a light blue tint, which makes them easier to see when handling.

### Lens Properties

· Refractive Index hydrated:

1.42

 Light Transmittance: . Oxygen Permeability (Dk): 93% (@ 610 nm, -1.000) 140 x 10<sup>-11</sup> (cm²/soc)(mi

Oz /ml x mm Hol. measured at 35° C (intrinsic Dk-Coulometric

method

· Water Content:

33% by weight in normal

saline

Surface Water Content:

≥ 80%

### Lens Parameters

13.0 to 15.0 mm Diameter Range

Spherical Power Range

-20.00 to +20.000

. Base Curve Range

8.0 to 9.2 mm

### Lens Parameters Available

### DAILIES TOTAL1\* (delefilcon A) spherical

Cherd Diameter:

14.1 mm

· Center Thickness:

0.09 mm @ -3.00D (varies

· Base Curve:

with power) 8.5 mm

· Powers:

-0.50 to -6.000 (0.250

steps); -6.50 to -12.000 (0.500 steps) +0.50 to +6.000 (0.250 steps)

### DAILIES TOTAL1\* Multifocal (delefficen A)

· Chord Diameter:

· Center Thickness:

0.09 mm @ -3.00D (varies

with power)

· Base Curve: Powers:

8.5 mm

+6,000 to -10,000 (0.250 steps) ADD: LO, MED, HI

NOTE: Hereafter, DAILIES TOTAL1\* spherical lenses and DAILIES TOTAL 1\* Multifocal contact lenses will simply be referred to as deleficon A contact lenses unless product distinction is necessary.

### ACTIONS

When hydrated and placed on the comea, defefficen A contact lenses act as a refracting medium to focus light rays on the retina.

### INDICATIONS (USES)

DAILIES TOTAL1\* (detefficion A) spherical soft contact lenses are Indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to approximately 1.50 diopters (D) of astigmalism that does not interfere with visual acuity.

DAILIES TOTAL1\* Multifocal (delefficon A) soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) and/or presbyopia in phakic or aphakic persons with non-diseased eyes who may require a reading addition of +3.00 (D) or less and who may have up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

The ienses are to be prescribed for single use, daily disposable wear. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

### **CONTRAINDICATIONS (REASONS NOT TO USE)** DO NOT use deletiicon A contact lenses when any of the following exists:

· Inflammation or infection of the anterior chamber of the eye

· Active disease, injury or abnormality affecting the comea, confunctiva, or evelide

- · Microbial infection of the eye
- Insufficiency of lacrimal secretion (dry eye) that Interferes with
- Corneal hypoesthesia (reduced corneal sensitivity)
- Use of any medication that is contraindicated or interferes with contact tens wear, including eye medications
   Any systemic disease which may be exacerbated by or
- interferes with contact lens wear
- · Allergic reactions or ocular imitation of the ocular surfaces or adnexa that may be caused by or exaggerated by the wearing of contact lenses
- Patient history of recurring eye or eyelid infections, adverse effects associated with contact lens wear, intolerance or abnormal ocular response to contact tens wear
- If eyes become red or irritated

Advise patients of the following warnings pertaining to contact

- · Problems with contact lenses and lens care products could result in serious injury to the eye. It is essential that patients follow their eye care professional's directions and all labeling Instructions for proper use of lenses and lens care products. Serious eye problems, including corneal ulcers, can develop rapidly and lead to loss of vision.
- Daily wear lenses are not indicated for overnight wear, and patients should be instructed not to wear lenses while sleeping. Clinical study results have shown that the risk of serious adverse reactions is increased when contact lanses are worn overnight?.
- Studies<sup>2</sup> have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than
- · If a patient experiences eye discomfort, foreign body sensation, estive tearing, vision changes, or redness of the eye, the patient should be instructed to immediately remove lenses and promptly contact his or her eye care professional. It is recommended that contact lens wearers see their eye care professional regularly as directed.

### **PRECAUTIONS**

To prevent damage to the eyes or to the contact lenses, the following precentions should be taken: Special Precentions for the Eye Care Professional: Due to the small number of patients enrolled in the clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated In significant numbers. Consequently when selecting an appropriate lens design and parameters, the eye care professional should consider all characteristics of the tens that can affect lens performance and ocular health, including oxygen permeability. central and peripheral thickness and optic zone diameter.
The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for retractive correction; therefore the continuing ocular health of the patient and lens performance on the aye should be carefully evaluated on initial dispensing and monitored on an ongoing basis by the prescribing eye care professional.

- Fluorescein, a yellow dye, should not be used while the lenses are on the patient's eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used, the eyes should be flushed thoroughly with sterile saline solution that is recommended for in eye use prior to inserting lenses. Avoid
- dispensing saline from an aerosol can directly into the eye. Patients who wear contact lenses to correct presbyopia may not achieve the best possible corrected visual aculty for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Before leaving the eye care professional's office, the patient should be able to promptly remove their lenses or should have someone else available who can remove their lenses for them. Eye care professionals should tristruct the patient to remove
- the lenses immediately if the eye becomes red or initiated.
- Routine eye examinations are necessary to help assure the continued health of the patient's eyes. Eye care professionals should make arrangements with the patient for appropriate

follow-up visits. Alcon recommends that patients see their eye care professional once each year, or more often, as recommended by the eye care professional.

Diabetics may have reduced comeal sensitivity and thus are

- more prone to comeal injury and do not heat as quickly or completely as non-diabetics.
- Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caudion patients

Eye Care Professionals should carefully instruct patients about the following safety precautions: Handling Precautions:

- Be sure that before leaving the eye care professional's office the patient is able to prompily remove lenses or have someone else available to remove them.
- Good hygiene habits help promote sale and comfortable lens wear. Always wash, rinse and thoroughly dry hands with a
- lint-free towel before handling lenses. REMOVE A LENS IMMEDIATELY if an eye becomes red or Inflated.
- Always handle lenses carefully. Never use tweezers or other sharp objects such as fingernalis to remove lenses from the iens container unless specifically indicated for that use.
- Do not use if blister package is damaged or not sealed completely. This may result in product contamination which can lead to a serious eye intection.
- Ensure that the correct lens for each eye is available. Shake the bilster pack gently prior to opening. Remove the lens from the bilster pack by carefully pouring the lens onto the palm of your clean hand. Ensure the lens is right side out, inspect lenses prior to insertion. Do not insert damaged lenses.
- To insert lenses:
  - Wash and rinse hands thoroughly and dry completely with a clean, fint free towel before handling tenses.
  - Place a lens on the tip of your clean and dry right or left index finger, place the middle finger of the same hand close to lower systashes and pull down the lower systle.

    Use the fingers of the other hand to lift the upper systle.

    Place the lens directly on the eye (cornea) and gently roll

  - finger away from the lens.
  - Look down and slowly remove the hand, releasing the lower lkd.
  - Look straight ahead and slowly remove the other hand, releasing the upper tid. - Blink gantly.
- To remove lenses:

  - Wash and rinse hands thoroughly and dry completely with a clean, lint free towel before handling lenses. Make sure hands are clean and completely dry. Blink fully several times.
  - While looking up, slide the lens down onto the white part of the eye.
  - Remove the lens by pinching gently between the thumb and forelinger. Do not pinch the eye tissue.
- If the lens is difficult to grasp, dry lingers once more and lry again. Do not use rewetting drops in this instance.
   If a lens decenters on the eye, it may be possible to recenter it.
  - Closing the eye and massaging the lens into piece, or
     Looking in the direction of the lens and blinking gently, or
  - Gently pushing the off-centered lens onto the comea with light finger pressure on the edge of the upper or lower
- eyelid.

  If a lens tears in the eye it will feel uncomfortable. Advise wearers it is impossible to lose a contact lens or part of a contact lens behind the eye and to remain calm. Lens pieces may be removed by plnching them as for normal lens removal, carefully avoiding pinching the eye tissue. If the tens pieces do not seem to remove easily, rinsing with saline is recommended. If this does not help, the wearer should contact an eye care professional for assistance.

### Lens Wearing Precautions:

- Patients should never exceed the prescribed wearing schedule regardless of how comfortable the lenses feet, Doing so may increase the risk of adverse effects.

  The lens should move freely on the eye at all times, if the lens
- the tens should move freely on the eye, to low the recommended directions in the Care for a Sticking Lens section. If non-movement of the lans continues, the patient should be instructed to consult their eye care professional immediately.

- The eye care professional should be consulted about wearing lenses during water sports and water related activities. Exposure to water or other non-sterile liquids while wearing contact lenses in activities such as swimming, water skiing, contact tenses in activities such as swimming, water sking, and hot tubs may increase the risk of octiar Intection, including but not limited to Acanthamoeba keralitis.

  Never allow contact lenses to come into contact with non-sterile liquids (including tap water and saliva) as microbial
- contamination can occur, which may lead to permanent eye
- trainings.

  Eye Inthation, Infection, or lens damage may result if cosmelics, totion, soap, cream, hair spray, deodorant, aerosol products or foreign particles come in contact with lenses.
- Environmental furnes, smoke, and vapore should be avoided in order to reduce the chance of tens contamination or physical trauma to the comea.
- · Lenses should be disposed of each day upon removal from the
- Discard any lens which has become dehydrated or damaged. Replace with a sterile, fresh, new lens.
- Note the correct lens power for each eye to prevent getting them mixed up.
- Always carry spare lenses with you or have back-up speciacles available.
- Do not share lenses with anyone as this may spread micro-organisms which could result in serious eye health problems
- · Do not use lenses beyond their expiration date.

### Other Topics to Discuss with Patients:

- Periodic eye examinations are extremely important for contact lens wearers. Schedule and conduct appropriate follow-up examinations to determine ocular response. Alcon recommends that patients see their eye care professional once
- each year or as recommended by the eye care professional once sach year or as recommended by the eye care professional. Certain medications may cause drynass of the eye, increased lens awareness, lens intolerance, and blurred vision or visual changes. These include, but are not limited to, antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness. Caution patients using such medications accordingly and prescribe proper remedial maasures.
- Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients

### Who Should Know that the Patlent is Wearing Contact Lenses:

- Pattenis should inform their health care practitioners that they are wearing contact lenses.
- Patients should inform their employers that they are wearing contact lenses. Some jobs may require the use of eye protection equipment or may require that contact lenses not be

It is strongly recommended that patients be provided with a copy of the DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal Contact Lenses (deleticon A) Patient instruction Booklet available from Alcon and understand its contents prior to dispensing the lenses.

### **ADVERSE EFFECTS**

Patients should be instructed to check eyes regularly to make sure they look well, feel comfortable and vision is clear. Potentially serious complications are usually accompanied by one or more of the following signs or symptoms:

Moderate to severe eye pain not relieved by removing the lens

- Foreign body sensation
- Excessive watering or other eye secretions including mucopurulent discharge
- Redness of the eyes
- Photophobia (light sensitivity)
- Burning, stinging or itching or other pain associated with the
- Comfort is less compared to when the lens was first placed on
- Poor visual acuity (reduced sharpness of vision)
   Blumed vision, rainbows or halos around objects
   Feeling of dryness

WHAT TO DO IF A PROBLEM OCCURS
Patients should be instructed that if any of the above signs or
symptoms are noticed, he or she should:

- IMMEDIATELY REMOVE THE LENSES.
- If the discomfort or problem stops, discard the lens and replace it with a new one.
- if the discomfort or problem continues after removing iens(es) or upon insertion of a new lens, IMMEDIATELY remove the lens(es) and contact the eye care professional for identification of the problem and prompt treatment to avoid serious eye damage.

  The patient should be informed that a serious condition
- such as corneal ulcer, infection, corneal vascularization, or

- idits may be present, and may progress rapidly. Less serious reactions such as abrasions, infiltrates, and bacterial conjunctivitis must be managed and treated carefully to avoid more serious complications.
- carefully to avoid more serious complications.
  Additionally, contact tens wear may be associated with ocular changes that require consideration of discontinuation or restriction of wear. These include but are not limited to local or generalized comeal adema, epithelial microcysts, epithelial staining, infiltrates, neovascularization, endothelial polymegathism, tarsal papillary changes, conjunctival injection

### **ADVERSE EFFECT REPORTING**

If a patient experiences any serious adverse effects associated with the use of DAILIES TOTAL 1\* brand (deletilcon A) contact lenses, please notify: Alcon Medical Safety in the USA at 1-800-757-9780.

### FITTING GUIDE AND PATIENT BOOKLET

Conventional methods of fitting contact lenses apply to delefficon A contact lenses. For a detailed description of the fitting techniques, refer to the DAILIES TOTAL1\* and DAILIES TOTAL1\* Multiflocal Contect Lenses (deleflicon A) Professional Fitting and Information Guide. Both the professional fitting guide and a patient instruction booklet are available free of charge from:

Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX, USA 76134-2099 1-800-241-5999

### LENS WEAR & REPLACEMENT SCHEDULES

- DAILY WEAH (less than 24 hours, while awake): To avoid tendency of the daily wear patient to overwear the
- To avoid tendency of the daily wear patient to overwear the
  lenses initially, stress the importance of adhering to a proper,
  initial wearing schedule. Normal daily wear of lenses assumes
  a minimum of 6 hours of non tens wear per 24 hour period.
   It may be advisable for patients who have never worn contact
  lenses previously to be given a wearing schedule that gradually
  increases wearing time over a few days. This allows more
  gradual adaptation of the ocular issues to contact lens wear.
- · The maximum daily wearing time should be determined by the eye care professional based upon the patient's physiological eye condition because individual responses to contact lenses vary. There may be a tendency for patients to overwear the lense initially. The eye care professional should stress the importance of adhering to the initial maximum wearing schedule. Studies have not been conducted to show schedule. Subject have not been consucred to snow that delefficin A contact lenses are safe to wear during sleep, therefore patients should be advised to remove their lenses while sleeping. Normal daily wear of lenses assumes a minimum of 6 hours of non-lens wear per 24 hour period. Optimum individual wearing schedule will vary.

  Detefficon A contact lenses are intended to be worn once (daily
- disposable wear) and then discarded at the end of each wearing period. The patient should be instructed to start the next wearing period with a fresh new lens.

### EMERGENCY LENS CARE

Cleaning and disinfection of daily disposable lenses is not recommended. The patient should be reminded to have replacement lenses or back-up speciacles available at all times.

### CARE FOR A STICKING LENS

If the tens sticks (stops moving) or begins to dry on the eye, instruct the patient to apply several drops of a recommended tubricating solution (used in accordance with package labeling). The palient should wait until the tens begins to move freely on the eys before attempting to remove it. It is important that the patient wash and dry their hands throroughly before removing the lens. If the lens continues to stick, the patient should IMMEDIATELY consult the eye care professional.

### IN OFFICE USE OF TRIAL LENSES

Eye care professionals should educate contact lens technicians concerning proper use of trial lenses.

Each contact lens is shipped sterile in a blister pack containing phosphate buffered saline solution. Hands should be thoroughly washed and rinsed saint sounds. Hards should be throughly washed and rinsed and dried with a lint-free towel prior to handling a lens. In order to ensure sterility, the bister pack should not be opened until immediately prior to use. For fitting and diagnostic purposes lenses should be disposed of after a single use and not be re-used from patient to patient.

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are epiashed into the eyes, the patient should:

Flush eyes immediately with tap water or fresh saline solution and immediately contact the eye care professional or visit a hospital emergency room without delay.

### **HOW SUPPLIED**

Each lens is packaged in a foli-sealed plastic container containing phosphate buttered saline solution with approximately 0.3% of phospharic currency some sound rains of opportunities of polyamic wetting agents consisting of copolymers of polyamidoamine and poly(cor)amide-acrylic) acid and is steam sterilized in the base curve, a sterilized in the base curve, and the steam of the diameter, dioptific power and ADD power (multifocal lenses), manufacturing tot number and expiration date.

### The following may appear on the labels or cartons:

| Symbols/Signs/<br>Abbreviations | Description |
|---|---|
| (Cont) | CAUTION: Federal hav (United States) restricts this device to sale by or on<br>the order of a licensed eye care professional. |
| STERRE | Steam sterifized |
| 2 60⊅ | Uso by date (Expiry date) |
| LOT | Batch code |
| <b>®</b> | Do not reuse |
| (6) | Do not use if blister package is demaged |
| <b>(D)</b> | Example of two letter language code (English) |
| DIA | Olameter |
| BC | Base curve |
| PWR | Power |
| D | Diopter (lens power) |
| ADD | Addition power |
| CEm | European conformity aign |
| $\Lambda$ | Caution |
| | See product instructions |
| <b>EE</b> | Authorized Representative European Community |
| | Manufacturer |
| 0 | Packeging waste license sign |

\* a trademark of Hovertis © 2016 Novertis

### Alcon Laboratories Inc.

6201 South Freeway Fort Worth, TX, USA 76134-2099 Www.alcon.com 1-800-241-5999

March 2016

W900038292-0316

Check for actual product availability as additional parameters may be

\*\*CRECK for Bettles produce systems as businesses personnectes step on introduced over time.

2 Schein, OD, Glynn RJ, Poggie EC, Seddon JM, Kenyon KR. The Relative Risk of Ulcerative Keratida Among Users of Daily Wear and Extended Wear Soft Contact lenses. H Eng J Med. 1989; 32321 (12;773-783)



### APPENDIX D: PRESBYOPIC SYMPTOMS QUESTIONNAIRE

Presbyopic Symptoms Questionnaire





### APPENDIX F: BINOCULAR OVER-REFRACTION

### APPENDIX G: BIOTRUE ONEDAY® FOR PRESBYOPIA FITTING GUIDE

### **BIOTRUE MULTI-FOCAL FITTING GUIDELINES**



### APPENDIX H: DAILIES TOTAL 1® MULTIFOCAL FITTING GUIDE

# Professional Fitting and Information Guide

DAILIES TOTAL1\*
and
DAILIES TOTAL1\* Multifocal
(delefilcon A) Soft Contact Lenses
For Single-Use, Daily Disposable Wear

**Water Gradient One-Day Contact Lenses** 



CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed eye care professional.



This page intentionally left blank

### **Table of Contents**

| Introduction | 5 |
|-----------------------------------------------------------|----|
| Product Description | 5 |
| Lens Properties | 6 |
| Available Lens Parameters | 6 |
| Actions | 6 |
| Indications (Uses) | 6 |
| Contraindications, Warnings, Precautions, Adverse Effects | 7 |
| Adverse Effect Reporting | 7 |
| Fitting Guidelines (Spherical Lenses) | 8 |
| Patient Selection | 8 |
| Pre-fitting Examination. | 8 |
| Trial Lens Evaluation | 8 |
| Lens Base Curve Selection | 8 |
| Initial Lens Power Selection | 8 |
| Lens Fit Assessment | 9 |
| Final Lens Power Determination | 10 |
| Fitting Guidelines (Multifocal Lenses) | 11 |
| Pre-Fitting Examination | 11 |
| Patient Selection | 11 |
| Initial Lens Selection | 13 |
| Initial Lens Fitting Evaluation | 14 |
| Initial Lens Visual Evaluation | 15 |
| Fitting Procedures | 16 |
| Fitting Guidelines (Monovision) | 18 |
| Patient Selection | 18 |
| Eye Selection | 18 |
| Special Fitting Considerations | 19 |
| Near Add Determination | 20 |
| Trial Lens Fitting | 20 |
| Adaptation | 20 |
| Other Suggestions | 21 |
| Dispensing Visit | 21 |
| Follow-Up Examinations | 23 |
| Follow-up Examination Procedures | 23 |
| Lens Handling Hints | 23 |
| Lens Insertion | 23 |
| Lens Removal | 24 |
| Care for a Sticking Lens | 25 |
| In Office Care of Trial Lenses | 25 |
| Additional information | 25 |
| Vertex Distance Conversion Chart | 29 |
| Product Package Insert | 29 |

This page intentionally left blank

### Introduction

Thank you for prescribing DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) daily disposable soft contact lenses. The benefits of a high oxygen transmissible and wettable lens material with a state of the art manufacturing process are combined to make DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) lenses. This guide contains important information regarding fitting procedures and aftercare of the DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) contact lens patient.

### **Daily Disposability:**

By eliminating the need for lens care, daily disposable lenses offer your patients a major advancement in wearing convenience. The next time you prescribe lenses consider the health and comfort benefits of beginning each wearing period with a new pair of fresh, sterile lenses that are worn once and then discarded.

### LightStream\* Lens Technology:

DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses are made from a proprietary silicone hydrogel material with a water content of approximately 33% water. The use of process automation, precision glass and quartz molds and photolithographic edge forming help ensure every lens has the same crisp optics, smooth surface finish and consistent edge quality from lens to lens. Delefilcon A contact lenses are produced under strictly controlled process conditions and inspected to exacting quality tolerances. As a result, you can be confident your patients will experience consistent vision, comfort, and ease of handling every day.

### **PRODUCT DESCRIPTION**

DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal soft contact lenses are made a silicone containing hydrogel that is approximately 33% water and 67% delefilcon A polymer with added phosphatidylcholine. The core lens material containing 33% water transitions through a water gradient to a hydrogel surface layer that exceeds 80% water. This structure enables a silicone hydrogel lens with a water gradient that has:

- Over 80% water at the surface of the lens to mimic the water content of the cornea.
- High level of oxygen transmissibility through the lens.
- Excellent overall comfort.

The lenses contain and release phosphatidylcholine (DMPC), a phospholipid found naturally in the tears. In addition, lenses contain the color additive copper phthalocyanine, a light blue tint which makes them easier to see when handling. The lenses are packaged in strips of 5 individual blisters containing buffered saline with approximately 0.3% of polymeric wetting agents consisting of copolymers of polyamidoamine and poly(acrylamide-acrylic acid).

### **Lens Properties**

Refractive Index (hydrated):

≥ 93% (@610 nm, -1.00D) Light Transmittance:

140 x 10<sup>-11</sup> (cm<sup>2</sup>/sec) Oxygen Permeability (Dk):

(ml O,/ml x mm Hg), measured at 35°C, (intrinsic Dk - Coulometric method)

Water Content 33% by weight in normal saline

Surface Water Content ≥ 80%

### Available Lens Parameters<sup>1</sup>

### DAILIES TOTAL1\* (delefilcon A) Spherical contact lenses

Chord Diameter Available: 14.1 mm

Center Thickness: 0.09 mm @ -3.00D (varies with power)

Base Curve: 8.5 mm

-0.50 to -6.00D (0.25D steps); -6.50 to Powers Available:

-12.00D (0.50D steps)

+0.50 to +6.00D (0.25D steps)

### DAILIES TOTAL1\* Multifocal (delefilcon A)

Chord Diameter: 14.1 mm

Center Thickness: 0.09 mm @ -3.00D (varies with power)

Base Curve: 8.5 mm

Powers: -0.25 to -10.00D (0.25D steps); plano to

+6.00D (0.25D steps) ADD: LO, MED, HI

<sup>1</sup>Check for actual product availability as additional parameters may be introduced over time.

### Actions

When hydrated and placed on the cornea delefilcon A soft contact lenses act as a refracting medium to focus light rays on the retina.

### **INDICATIONS (USES)**

DAILIES TOTAL1\* (delefilcon A) spherical soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) and/or presbyopia in phakic or aphakic persons with non-diseased eyes who may require a reading addition of +3.00 (D) or less and who may have up to approximately 1,50 diopters (D) of astigmatism that does not interfere with visual acuity.

The lenses are to be prescribed for single use, daily disposable wear. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

See WARNINGS for information about the relationship between wearing schedule and corneal complications.

### CONTRAINDICATIONS, WARNINGS, PRECAUTIONS AND ADVERSE EFFECTS

For additional important prescribing and safety information, refer to the Package Insert that is printed in the back of this guide.

### ADVERSE EFFECT REPORTING

If a patient experiences any serious adverse effects associated with the use of DAILIES TOTAL1\* or DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses, in the USA please contact Alcon Medical Safety at 1-800-757-9780.

### **FITTING GUIDELINES**

Please see the appropriate sections of this booklet that contain guidelines for spherical, multifocal and monovision fitting techniques.

### **FITTING GUIDELINES (Spherical Lenses)**

### 1. Patient Selection

The patient characteristics necessary to achieve success with DAILIES TOTAL1\* (delefilcon A) spherical lenses are similar to those for other spherical soft contact lenses. A thorough pre-fitting examination should be conducted to ensure the patient is a suitable candidate for soft contact lens wear.

The following procedures should be followed when fitting DAILIES TOTAL1\* (delefilcon A) spherical lenses. For additional tips on fitting the monovision patient refer to the section *Monovision Fitting Guidelines*.

### 2. Pre-fitting Examination

### A pre-fitting examination is necessary to:

- assess the patient's motivation, physical state and willingness to comply with instructions regarding hygiene and wear schedule
- make ocular measurements for initial contact lens parameter selection
- collect baseline clinical information to which post-fitting examination results can be compared

### A pre-fitting examination should include:

- a thorough case history
- · a spherocylindrical refraction
- keratometry
- tear film assessment
- biomicroscopy

### 3. Trial Lens Evaluation

### A. Lens Base Curve Selection

A well-fitted lens provides good movement, centration and comfort. An optimal fit can be achieved for the vast majority of patients with the single 8.5 mm base curve.

### B. Initial Lens Power Selection

The initial power selection should be as close as possible to the patient's prescription after taking into account spherical equivalent and vertex calculations, if necessary.

### Spherical Equivalent Calculation

To determine initial lens power, convert the spherocylindrical spectacle Rx to its spherical equivalent as follows:

Spherical Equivalent = Sphere power + 1/2 (Cylinder Power)
Example: Spectacle Rx: -4.50D -1.00 x 180

Spherical equivalent: -4.50D + (-0.50D) = -5.00D

### **Vertex Distance Conversion**

If the spherical equivalent is greater than  $\pm$  4.00D, a vertex distance correction is necessary (see *Vertex Distance Conversion Chart*) to determine the lens power required at the corneal plane.

Example:

Spectacle Rx:

-4.50D -1.00 x 180

Spherical equivalent:

-4.50D + (-0.50D) = -5.00D

Vertex compensation:

-4.75 (initial lens power)

### C. Lens Fit Assessment

Allow the lenses to settle on the eyes for approximately 10 minutes. This allows time for the patient to adapt to the lenses and time for the lens to equilibrate.

Evaluate the fit and movement of the lenses on the eye in primary and up gaze positions. The **Push-up Test**, as described below, is an additional test of the lens evaluation. The following guidelines will be helpful in fit evaluation:

### Characteristics of a Well-fitted Lens

A well-fitted DAILIES TOTAL1\* (delefilcon A) spherical contact lens satisfies the following criteria:

- 1. Good centration and full corneal coverage in all fields of gaze.
- Sufficient lens movement to allow tear exchange under the lens during a blink in primary or upward gaze.
- 3. Satisfactory Push-up Test
  - This test is a reliable indicator of a good fit. With the patient looking straight ahead, place your index finger on the patient's lower lid and nudge the edge of the lens upward while observing lens movement. Then pull the lid back down and observe the return of the lens.
  - A well fitted lens will move freely upward, stopping shortly after passing the limbus and then return freely to its original position.
- Good comfort and stable visual response (with over refraction).

### Characteristics of a Tight (Steep) Lens Fit

A tight or steep lens fit would display some or all of the following characteristics:

- Insufficient or no lens movement during a blink in primary or upward gaze.
- 2. Unsatisfactory Push-up Test
  - A tight fitting lens will resist movement. If successfully nudged upward, the lens may remain decentered or return slowly to its original position.
- 3. Good centration.
- 4. Good comfort.
- 5. Fluctuating vision between blinks.

### Characteristics of a Loose (Flat) Lens Fit

A loose lens fit would display some or all of the following characteristics:

- 1. Reduced comfort, usually accompanied by lower lid sensation.
- Poor centration with limbal exposure on exaggerated eye movement.
- 3. Lens edge standoff.
- 4. Excessive iens movement during the blink in primary or upward
- 5. Unsatisfactory Push-up Test
  - A loose fitting lens will move easily but may remain decentered or slip under the upper lid.
- 6. Vision may be blurred after the blink.

An inverted lens may mimic the characteristics of a loose lens. If any of

the above signs occur remove the lens and check to make sure it is not inverted.

### **General Fitting Tips**

- Trial fitting of the individual eye is recommended.
  A well fitting lens will show movement of 0.1 to 0.5 mm.
  Final Lens Power Determination

After the characteristics of a well fitted lens have been satisfied, conduct a spherical over-refraction to determine the proper lens power to be dispensed.

Example:

Diagnostic lens: Over-refraction:

-4.50 -0.25

Final lens power:

-4.75

### FITTING GUIDELINES (Multifocal)

The DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lens is a progressive aspheric simultaneous vision soft contact lens, intended to correct presbyopia with or without additional ammetropia, available in three ADD powers; low (LO), medium (MED) and high (HI). For each lens the near and intermediate powers are concentrated primarily in the central portion of the optical zone while the distance power is contained in the surrounding portion. The continuous changes in power across the surface of the lens allow patients requiring a reading addition of up to + 3.00D to see clearly at far, intermediate, and near distances.

Achieving high success with DAILIES TOTAL1\* Multifocal (deleficon A) contact lenses is dependent on several factors, including the patient's motivation, expectations and visual wearing environment, as well as your skill in optimizing the lens powers to balance binocular performance at distance and near. The information in this guide is designed to provide you with the tools to manage your presbyopic patients through each stage of the process from the initial case history to post-fitting follow-up.

### 1. Pre-fitting Examination

### A pre-fitting examination is necessary to:

- determine whether a patient is a suitable candidate for DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses
- make ocular measurements and assessments for initial contact lens parameter selection
- collect baseline clinical information to which post-fitting examination results can be compared

### A pre-fitting examination should include:

- a thorough case history
- detailed assessment of patient's individual visual demands
- understanding of patient's objectives for lens wear and expectations
- a distance spherocylindrical refraction, near add determination and measurement of pupil diameter
- keratometry
- · tear assessment
- biomicroscopy

Note: The importance of a thorough case history should not be underestimated. The information gained through careful listening and probing will help greatly in satisfying each patient's unique needs.

### 2. Patient Selection

The eye care professional should weigh several factors when considering patient selection for a DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lens fitting. When fitting a lens intended to correct for presbyopia, it is especially important to evaluate the particular visual needs, objectives, lifestyle and expectations of the individual patient. Prospective candidates may include current contact lens wearers, former wearers, and persons with no previous wear history. For former wearers it is important to determine the cause for discontinuation.

There are two general categories of candidates based on anticipated usage: those who seek to wear their lenses as their principal means

of vision correction, and those who wish to integrate the use of their contact lenses with spectacles. The integrative user often seeks to wear their lenses for sports or other occasional activities while reverting to spectacles under poor lighting or otherwise demanding vision conditions. In general, even the part-time user does not require more than a few moments re-adaptation time following an interval of no lens wear.

While candidates with greater than 1.00 diopter of refractive error have often been thought of as better candidates than those with low error or emmetropia, this is a generalization that often does not hold true for a given individual. Success is influenced by many factors and the eye care professional is encouraged to offer DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses to all interested presbyopic patients who satisfy the standard requirements for soft contact lens wear.

To summarize patient selection, the characteristics of "ideal candidates" and those that will be more difficult to fit" are listed below:

### Ideal Candidates

- Refractive cylinder < 1.00D.</li>
- Attainable visual demands that do not depend upon resolving very fine (smaller than 20/20 letters) details at both distance and near for extended periods while wearing DAILIES TOTAL1\* Multifocal contact lenses.
- Emphasis on tasks where it is advantageous to have objects simultaneously in focus over a large range of viewing distances.
- Expectations consistent with actual everyday visual demands.
- Motivated to wear lenses and understands that vision may not always be as sharp as with spectacles for some distances or lighting conditions.
- Unable to adapt to monovision correction.

### Less than Ideal Candidates

- Critical or very fine visual demands at both distance and near.
- Refractive cylinder ≥ 1.00D (any axis) in one or both eyes or against-the-rule refractive cylinder > 1.00D in one or both eyes.
- Monocular distance acuities poorer than 20/20 with spherical equivalent refractive correction.
- Myopic anisometropia where the refractive error for one of the two eyes is low (≤1.50D) and has not been habitually corrected.
- Pupil size larger (> 4 mm) or smaller (<3 mm) than norm for presbyopic population under natural illumination conditions.
- Abnormal binocular sensory function (e.g., amblyopia or strabismus).
- Expectation to discard and never use spectacles again, including reading glasses, even for special tasks or viewing conditions.
- Highly satisfied monovision wearers.
- Any other contraindications to successful contact lens wear such as tear abnormality or lid margin disease.

### 3. Initial Lens Selection

A. Initial Base Curve Selection

DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses are available in a single 8.5 mm base curve.

### B. Initial Lens Power Selection

Note: A careful maximum plus spherocylindrical refraction and nearpoint add determination should be conducted prior to selecting a DAILIES TOTAL1\* Multifocal (delefilcon A) trial lens. Autorefraction findings should be refined manually to rule out effects of instrument myopia and ensure proper control of residual accommodation.

The DAILIES TOTAL1\* Multifocal lens design makes selecting the initial lens power easy. You need only manipulate the distance power. The optimum starting point is with a power that is equal to or more plus or less minus than the vertex corrected spherical equivalent spectacle refraction.

### C. Initial ADD Selection

Note: A careful nearpoint ADD determination should be conducted prior to selecting a DAILIES TOTAL1\* Multifocal (delefilcon A) trial lens

The DAILIES TOTAL1\* Multifocal (delefilcon A) 3 ADD SYSTEM allows personalized fitting for presbyopic patients. The table below makes initial ADD selection easy.

### DAILIES TOTAL1\* MULTIFOCAL ADD SELECTION

| SPECTACLE ADD | BOTH EYES |
|----------------|------------|
| Up to +1.25 | © |
| +1.50 to +2.00 | <b>(</b> |
| +2.25 to +2.50 | <b>(b)</b> |

| Example 1: | OD | | OS |
|-------------------------------------|------------------|--------|----------|
| Spherical Rx: | -4.50 -0.75 x 90 | | -4.00D |
| Spherical equivalent (least minus); | -4.75D | | -4.00D |
| Vertex corrected power: | -4.50D | | -4.00D |
| Spectacle Add: | | +0.75D | |
| Eye Dominance: | | OD | |
| Initial Trial Lens: | -4.50 LO | | -4.00 LO |

| Example 2: | OD | | os |
|---|---|---|---|
| Spherical Rx: | +4.25 -0.25 x 180 | | +4.00 D<br>-0.50 x 180 |
| Spherical equivalent (least minus): | +4.25D | | +3.75D |
| Vertex corrected power: | +4.50D | | +3.75D |
| Spectacle Add: | | +2.00D | |
| Eye Dominance: | | os | |
| initial Trial Lens: | +4.50 MED | | +3.75 MED |

### 4. Initial Lens Fitting Evaluation

- a) Insert the lenses selected in Section 3 (above). If the exact power is not available, choose the next closest least minus/most plus lens power in your trial set.
- b) Allow the lenses to settle on the eyes for approximately 10 minutes. This allows time for the patient to adapt to the lenses and time for the lens to equilibrate with the patient's tears.
- c) Evaluate the fit of the lenses on the eye. The Push-up Test as described below is an important part of the lens evaluation. The following guidelines will be helpful in evaluating the physical fit of the lens:

### Characteristics of a Well-fitted Lens

A well-fitted DAILIES TOTAL1\* Multifocal (delefilcon A) contact lens satisfies the following criteria:

- Full corneal coverage and good centration (no limbal exposure).
   A lens that is decentered > 1 mm, particularly temporal, is less likely to give adequate vision.
- Lens movement of 0.1 to 0.5 mm should be present to allow tear exchange under the lens during a blink in primary gaze or upward gaze and to avoid variable vision.

### **Push-up Test:**

- This test is a reliable indicator of a good fit. With the patient looking straight ahead, place your index finger on the patient's lower lid and nudge the edge of the lens upward while observing lens movement. Then puil the lid back down and observe the return of the lens.
- A well fitted lens will move freely upward, stopping shortly after passing the limbus and then return freely to its original position.
- 3. Good comfort.
- 4. Acceptable visual acuity with over-refraction.

### Characteristics of a Tight (Steep) Lens Fit

A tight or steep fit should not be dispensed. If a lens fit is judged to be too steep a flatter lens (larger base curve), if available, should be evaluated. A tight or steep lens fit would display some or all of the following characteristics:

- 1. Good centration.
- Insufficient or no lens movement during a blink in primary gaze or upward gaze.
- 3. Excessive conjunctival drag (visible movement of the conjunctival vessels when the lens moves during a blink or during the push-up test). Note: presbyopes often have loose conjunctiva, some conjunctival movement is occasionally seen and may not be a sign of a tight fit. See Push-up Test below.

  Push-up Test:
  - A tight fitting lens will resist movement. If successfully nudged upward, the lens may remain decentered or return slowly to its original position.
- 4. Good comfort.
- 5. Blurred vision between blinks.

### Characteristics of a Loose (Flat) Lens Fit

If a lens fit is judged to be too flat a steeper lens (smaller base curve), if available, should be evaluated. A loose lens fit would display some or all of the following characteristics:

- 1. Decentration.
- Excessive lens movement during the blink in primary or upward gaze.

### Push-up Test:

- A loose fitting lens will move very easily, well beyond the limbus and possibly encroaching upon or going beyond the pupil. It will then return very quickly to its original position and often times return lower than its original position.
- 3. Reduced comfort.
- 4. Lens edge standoff.
- 5. Blurred vision immediately after the blink.

### 5. Initial Lens Visual Evaluation

While lenses are settling, it is helpful to take the patient from the exam room to a "real-world" setting such as a room with an outside view. Once an acceptable fit has been achieved, the visual performance of the lenses may be evaluated. Visual acuity is tested at distance. If necessary, a spherical over-refraction should be performed using a trial frame or hand held lenses rather than a phoropter. This technique is essential when fitting multifocal lenses because it allows the patient to maintain the head posture and direction of gaze (relationship between eye and head) that he or she would naturally use during everyday tasks. This ensures that the visual performance of the lens is being assessed under conditions where the on-eye positioning matches that which will occur when the lens is being used, for example, for near work activities. In addition, pupil size will not be artificially increased

by the reduction in light associated with looking through the aperture of the phoropter cells, or decreased by proximal cues associated with the nearness of the instrument.

### 6. Fitting Procedures

Step 1. After the trial lenses have settled for approximately 10 minutes, measure distance acuity while the patient is viewing the chart binocularly (i.e., simultaneously with both eyes). Next, evaluate the patient's subjective impression of the near vision when trying to read typical everyday material (e.g., a newspaper, magazine, and cell phone). Lighting and reading distance should be what is normal for the patient.

Step 2. If distance or near vision is unsatisfactory, perform a binocular distance over-refraction, as follows. Use hand-held trial lenses and encourage plus. For example, if a Plano and +0.25D over-refraction yields the same results, use the +0.25D endpoint. Re-check visual acuity and visual quality as described in Step 1 above. If over-refraction is other than plano, go immediately to new trial lenses, keeping ADD the same.

Step 3. If distance and near vision are satisfactory, dispense lenses and remind patient to use good light when reading fine print or use additional reading glasses if needed. It is helpful to let the patient experience the lenses in their natural environment before further procedures for enhancing vision are performed.

Step 4. Enhanced Near Vision. If near vision is unsatisfactory, determine the dominant eye by the following method. Determine the eye with greatest plus acceptance by placing +1.50 handheld trial lens over each eye alternately while patient views in the distance with both eyes open. Consider the eye for which binocular vision blurs *least* with the +1.50 to be the non-dominant eye. Other methods to determine the dominant eye are appropriate.

Step 4A: Check the patient's binocular acuity with +0.50 over the non-dominant eye to determine if near vision is improved and distance vision is still acceptable. If so, place a new trial lens with the same ADD on the non-dominant eye, adjusting the distance power by +0.50.

| Enhanced near vision, Step A | | |
|---|---|---|
| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT EYE<br>(PLUS ACCEPTED) |
| Up to +1.25 | 6 | with additional +0.50 |
| +1.50 to +2.00 | (dia) | with additional +0.50 |
| +2.25 to +2.50 | • | with additional +0.50 |

Next, re-check visual acuity and visual quality as described in Step 1 above. If satisfactory, dispense new distance lens power for the non-dominant eye. If near vision is still unsatisfactory, proceed to Step B:

Step 4B: If near vision is still unsatisfactory, adjust ADD as shown below.

| Enhanced near vision, Step B | | |
|---|---|---|
| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT EYE<br>(PLUS ACCEPTED) |
| Up to +1.25 | 4 | <b>(</b> 1) |
| +1.50 to +2.00 | <b>(3)</b> | 6 |
| +2.25 to +2.50 | • | - 6 |

Note: It is common to question the rather non-intuitive step we suggest for enhancing vision at near in the HI ADD range, where the suggestion is to "back off" to a MED ADD for the non-dominant eye, the same suggestion we make for enhancing distance vision (below). The reason for this is that after establishing (in Step A) that increasing plus is not helpful, the next most common reason for blur at near (or distance) is unacceptable ghosting that degrades the image quality. Backing down to the MED ADD in one eye can often relieve that and actually improve vision at near.

<u>Step 5</u>: Enhanced Distance Vision. If distance over-refraction did not improve visual acuity, adjust ADD according to the chart below.

| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT<br>EYE<br>(PLUS ACCEPTED) |
|----------------|--------------|----------------------------------------|
| +1.50 to +2.00 | 0 | <b>(40)</b> |
| +2.25 to +2.50 | Ð | (in) |

### FITTING GUIDELINES (Monovision) Patient Selection

### A. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. Patients with reduced visual acuity, such as the amblyopic patient, may not be a good candidate for monovision.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it must be determined by trial whether this patient can function adequately with monovision. Monovision contact lens wear may not be optimal for such activities as:

- visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- driving automobiles (e.g., driving at night). Patients who cannot
  pass requirements for a driver's license with monovision
  correction should not drive with this correction. An additional
  over-correction can be prescribed to improve vision.

### B. Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with bifocal reading glasses. Each patient must understand that monovision, as well as other presbyopic contact lenses, or other alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision in straight-ahead and upward gaze that monovision contact lenses provide compared to spectacle bifocals.

### **Eye Selection**

Generally, the non-dominant eye is corrected for near vision. The following test for eye dominance can be used:

### A). Ocular Preference Determination Methods

- Method 1 Determine which eye is the "sight eye". Have the
  patient point to an object at the far end of the room. Cover
  one eye. If the patient is still pointing directly at the object,
  the eye being used is the dominant (sighting) eye.
- Method 2 Determine which eye will accept the added power for near with the least reduction in distance vision. Place a trial spectacle near ADD lens in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

### B). Refractive Error Method

 For anisometropic corrections, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near. C). Visual Demands Method

 Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

Example:

A person who places copy to the left side of the desk will usually function best with the near lens on the left eye.

### **Special Fitting Considerations**

Unitateral Lens Correction

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens while a bilateral myope may require only a distance lens.

Examples:

 Emmetrope: A presbyopic emmetropic patient who requires a +1.75 diopter ADD would have a +1.75 lens on the near eye and the other eye left without a lens.

 Bilateral myope: A presbyopic patient requiring a +1.50 diopter ADD who is -2.50 diopters myopic in the right eye and -1.50 diopters myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.

Unllateral astigmat:

a) Emmetropic in one eye, astigmatic in the other

Spectacle Rx
O.D. Plano
O.S. -1.00 -1.00 x 090
Add: +1.50

Potential Monovision Rx
Uncorrected for distance
+0.50 -1.00 x 090 for near

b) Myopic in one eye, astigmatic in the other

Ambiyopia

The amblyopic patient may not be a good candidate for monovision. Astigmatism

Patients with less than 1.50 diopters of astigmatism might be successfully fit in DAILIES TOTAL1\* (delefilcon A) spherical lenses.

- Determine which eye to use for the near prescription (see Eye Selection, A-C, above)
- Add the appropriate near add power to the spherical component of the astigmatic prescription for that eye.

| Example: | Spectacle Rx | Potential Monovision Rx |
|----------|-------------------------|--------------------------------|
| | O.D.: -2.50 -0.75 x 180 | -2.50 -0.75 x 180 for distance |
| | O.S.: -3.00 -1.75 x 165 | -2.00 -1.75 x 165 for near |
| | Add: +1.00 | |
| | Dominant eye: O.D. | |

### **Near Add Determination**

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

### **Trial Lens Fitting**

A trial lens fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the directions in the *General Fitting Guidelines and Base Curve Selection* described earlier in the guide.

Case history and standard clinical evaluation procedures should be used to determine the suitability of monovision. Determine which eye is to be corrected for distance and which eye is to be corrected for near. Next determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Immediately after the correct power lenses are in place, walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tasks are completed, should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to news print and finally smaller type sizes.

After evaluating the patient's performance under the above conditions, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a less favorable prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

### Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a few minutes or for several weeks. The longer these symptoms persist, the poorer the chance for successful adaptation. To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it is recommended that patients be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several

weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive under optimal driving conditions. After adaptation, and success with these activities, the patient should be able to drive under other conditions with caution.

**Other Suggestions** 

The success of the monovision technique may be further improved by having your patient follow the suggestions below:

 Have a third contact lens (distance power) to use when critical distance viewing is needed.

 Have a third contact lens (near power) to use when critical near viewing is needed.

- Have supplemental spectacles to wear over the monovision contact lenses for specific visual tasks. This is particularly applicable for those patients who cannot meet driver's licensing requirements with a monovision correction.
- Make use of proper illumination when carrying out visual tasks.

Success in fitting monovision can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of the clear near vision in straight ahead and upward gaze with monovision.

The decision to fit a patient with a monovision correction is most appropriately left to the eye care professional in conjunction with the patient after carefully considering the patient's needs. All patients should be supplied with a copy of the Patient Instruction Booklet, which contains important instructions for the monovision wearer. You can obtain copies of the instruction book by calling customer service in the USA at (800) 241-5999.

### **DISPENSING VISIT**

To help ensure patient success the following steps should be conducted with each patient, even if they have previously worn contact lenses. Even experienced wearers are prone to develop bad habits over time.

DAILIES TOTAL1\* brand (delefilcon A) lenses are supplied sterile in foil sealed blister pack containers. Open the foil pack by peeling back the foil lidding material and gently slide the lens out of the container with your finger, or pour the lens onto the palm of your clean hand.

Conduct the following steps with each patient, even if they have previously worn contact lenses:

### A. Verification of Lens Fit

Evaluate lens fit and visual response with the lens on the eye. The criteria of a well-fitted lens should be met and the patient's visual acuity should be acceptable. If not, the patient should be refitted with a more appropriate lens.

### B. Hygiene and Lens Handling Instructions

Good hygiene and proper lens handling are important factors in achieving safe, comfortable lens wear. Instruct the patient on hygiene and handling of lenses. Patients who are unable to place and remove lenses should not be provided with them.

### C. Lens Wear and Replacement Schedules (see Package Insert)

Prescribe and explain the daily disposable wear schedule. Explain that lenses are to be discarded after each daily wearing period. Determine the maximum suggested daily wearing period based on the patient's physiological eye condition. There may be a tendency for the patient to overwear their lenses initially. For some patients who have never worn contact lenses consider a wearing schedule that allows for a gradual increase in wearing time.

### D. Lens Care Directions (see Package Insert)

The lenses are not intended to be cleaned or disinfected and should be discarded after a single use. The eye care professional may recommend lens rewetting drops, as needed.

### E. Specific Instructions for Presbyopic Patients

Specific instructions, explanations and demonstrations are important for optimizing patient success with multifocal contact lenses. The following information and instructions have proven useful in advising patients who wear DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lenses.

- A contact lens that contains different powers for distance and near involves greater technological and optical complexity than does a bifocal or multifocal spectacle lens. This is because the contact lens moves with the eye, rather than having the eye move up and down while the lens remains suspended in a frame. While the contact lens therefore gives an unobstructed field of view and greater freedom regarding where to look, these advantages may mean that the sharpness of vision may not always be exactly the same as what would be experienced with spectacles.
- Although many individuals use DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses for full-time wear, it is not unusual to find that there may be some activities where one prefers to wear spectacles, or where the disadvantages associated with spectacles are outweighed by other issues. This is an entirely normal and natural response to the challenges presented by presbyopia.
- Situations where vision with multifocal contact lenses may be less sharp or otherwise "different" than what is experienced with spectacles often involve low illumination (e.g., a semi-dark room), reduced visibility (e.g., outdoor conditions of fog or heavy rain), or isolated sources of very bright light (e.g., headlights of an oncoming vehicle on a narrow country road). Patients should be instructed to make use of good light when reading fine print.
- Patients should be aware that it might be advisable to refrain from wearing their lenses while driving, flying an airplane or operating heavy machinery while wearing their lenses until they gain some experience with the lenses in a similar visual environment.
- Small changes in lens power can often make a significant difference in the quality of the vision experienced with multifocal contact lenses. Such changes can be best tailored to

individual needs and environmental conditions that the patient will personally encounter on a day-to-day basis. Confidence and assurance that such refinements, if needed, can be achieved are important for patient motivation during the initial period of lens wear.

### F. Additional Instructions

Review the Package Insert

Provide the patient with all relevant information and precautions on

the proper use of the lenses that are prescribed.

Provide the Patient Instruction Booklet for DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefficon A) Contact Lenses. Give the patient a copy of the Patient Instruction Booklet for DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lenses. Review the contents so the patient clearly understands the prescribed lens wear, care, and replacement schedule. In the USA you can obtain copies of the instruction book by calling Alcon customer service at (800) 241-5999.

### Follow-Up Examinations

Follow-up care is extremely important for continued successful contact lens wear. Follow-up care should include:

- Case history, including questions to identify any problems related to contact lens wear
- Management of specific problems, if any, and
- A review with the patient of the lens wearing schedule, replacement schedule and handling procedures.

### Follow-up Examination Procedures

- Patients should be instructed to wear lenses prior to a follow-up examination.
- Record patient's symptoms, if any.
- Measure visual acuity monocularly and binocularly with the contact lenses in place.
- Perform an over-refraction to check for residual refractive error.
- With a biomicroscope, evaluate lens fitting.
- Remove the lenses and conduct a thorough biomicroscopic examination with fluorescein. Rinse eyes with saline before re-inserting lenses.
- Evert upper lids to determine condition of tarsal conjunctiva.
- Periodically perform keratometry and spectacle refractions. These results should be recorded to compare to the initial measurements.
- If any observations are abnormal, use professional judgment to manage the problem and restore the eye to optimal conditions. If visual requirements are not satisfied during any follow-up examination, the patient should be re-fitted with a more appropriate lens.

### **LENS HANDLING HINTS**

### Lens Insertion

When about to place the lens on the eye, make sure the lens sits up on the placement finger. The finger should be dry so surface tension does

not cause the lens to adhere to the finger.

 Check to see that the lens is right side out. A lens that is placed on the eye inside out may not feel comfortable or provide good vision.

One way to do this is to perform the 'taco test' by placing the lens between your thumb and index finger and squeeze the edges together gently.

If the edges come together, the lens is right side out.

 If the edges turn outward, the lens is wrong side out. Carefully reverse it with your fingers.



Another way is to place the lens on the tip of your index finger and check its shape.

If the edge appears bowl-shaped, it is right side out.

- If the edge has a lip or flares outward, it is wrong side out and must be reversed.
- Place the lens directly onto the comea (placing it on the lower sclera can lead to the lens folding after a blink). While continuing to hold both lids in place, the patient should look down to seat the lens. The lids may then be released.



### Lens Removal

- Wash hands thoroughly with soap that does not have any oils, lotions or perfumes.
- · Carefully dry hands with a clean, lint-free towel.

It is important to remind patients to dry their hands thoroughly prior to removing their lenses. The surface of DAILIES TOTAL1\* brand lenses is designed to stay very wet and lubricious, or slippery while on the eye. If their fingertips are wet they are likely to slip across the surface of the lens making removal more difficult.

- Slide the lens off the cornea (down or to the side) onto the sclera. This
  produces a fold in the lens, which assists in removal. With the index finger
  and thumb, gently pinch the lens off the eye.
- Discard lenses.
Care for a Sticking Lens

• In the unlikely event that the lens sticks (stops moving) or begins to dry on the eye, instruct the patient to apply several drops of a recommended lubricating solution (used in accordance with package labeling). The patient should wait until the lens begins to move freely on the eye before attempting to remove it. If the lens continues to stick, the patient should immediately consult the eye care professional.

#### IN OFFICE CARE OF TRIAL LENSES

Eye care professionals should understand and educate contact lens technicians concerning proper use of trial lenses.

Each contact lens is shipped sterile in a sealed blister pack containing phosphate buffered saline with additives. Hands should be thoroughly washed and rinsed and dried with a lint-free towel prior to handling a lens. In order to insure sterility, the blister pack should not be opened until immediately prior to use.

 Delefilcon A lenses are for daily disposable wear only and should be discarded after a single use. The lenses should be disposed of after a single use and not be re-used from patient to patient.

#### ADDITIONAL INFORMATION

For assistance with fitting or clinical questions regarding DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal contact lenses eye care professionals having questions or problems should contact Medical Information Systems in the USA at (800) 241-7468. To order DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal contact lenses contact your Alcon sales representative or call Customer Service, in the USA at (800) 241-5999.

#### **VERTEX DISTANCE CONVERSION CHART**

For minus lenses, read left to right; for plus lenses, read right to left. (12 mm Vertex Distance)

| * | + | * | + | * | + | ew . | + |
|------|------|-------|-------|-------|-------|-------|-------|
| 4.00 | 3.87 | 7.50 | 6.87 | 12.00 | 10.37 | 19.00 | 15.50 |
| 4.25 | 4.00 | 7.62 | 7.00 | 12.50 | 10.75 | 19.25 | 15.62 |
| 4.50 | 4.25 | 7.75 | 7.12 | 12.75 | 11.00 | 19.25 | 15.75 |
| 4.75 | 4.50 | 7.87 | 7.25 | 13.00 | 11.25 | 19.75 | 16.00 |
| 5.00 | 4.75 | 8.00 | 7.37 | 13.50 | 11.50 | 20.00 | 16.12 |
| 5.12 | 4.87 | 8.12 | 7.50 | 13.75 | 11.75 | 20.25 | 16.25 |
| 5.37 | 5.00 | 8.25 | 7.62 | 14.00 | 12.00 | 20.50 | 16.50 |
| 5.50 | 5.12 | 8.50 | 7.75 | 14.25 | 12.25 | 20.75 | 16.62 |
| 5.62 | 5.25 | 8.75 | 8.00 | 14.75 | 12.50 | 21.00 | 16.75 |
| 5.75 | 5.37 | 9.00 | 8.25 | 15.00 | 12.75 | 21.25 | 17.00 |
| 5.87 | 5.50 | 9.25 | 8.37 | 15.50 | 12.75 | 21.75 | 17.25 |
| 6.00 | 5.62 | 9.50 | 8.62 | 15.75 | 13.25 | 22.25 | 17.50 |
| 6.12 | 5.75 | 9.75 | 8.75 | 16.25 | 13.50 | 22.50 | 17.75 |
| 6.37 | 5.87 | 10.00 | 9.00 | 16.75 | 13.75 | 23.00 | 18.00 |
| 6.50 | 6.00 | 10.25 | 9.12 | 17.00 | 14.00 | 23.50 | 18.25 |
| 6.62 | 6.12 | 10.50 | 9.25 | 17.25 | 14.25 | 23.75 | 18.50 |
| 6.75 | 6.25 | 10.75 | 9.37 | 17.62 | 14.37 | 24.25 | 18.75 |
| 6.87 | 6.37 | 11.00 | 9.62 | 18.00 | 14.50 | 24.75 | 19.00 |
| 7.00 | 6.50 | 11.25 | 9.75 | 18.12 | 14.75 | 25.00 | 19.25 |
| 7.12 | 6.62 | 11.50 | 10.00 | 18.50 | 15.00 | 25.50 | 19.50 |
| 7.37 | 6.75 | 11.75 | 10.25 | 18.75 | 15.25 | 26.00 | 19.75 |

This page intentionally left blank

Barterians fine persons count a efection and sharen first and apply and to be object in account to love, these accounts below, these materials and inceptor orientation for himse and, first personal or any processed, but death to encode a country to proceed a country to the co

(I) only

PHOCOUT DESCRIPTION
SMR.RE THTAL1" and DAR RE THTAL1" Multiforal fedical Re-selt confect branes are made from a lone material and in 22% priest and 67% fedicificat Alphymes, a alloans containing

| tyringel selb arten programicy<br>contribute 11% under benedere<br>tyringel autace byer that proper<br>color additive copper philistocyan<br>than earlier to see when knocking | Busugh & maler gradient to a<br>la BOX busige, Leonar contain th<br>ire, a light bile tint, which make |
|---|---|
| Law Proporties | |
| · Retractiva frater bydratud. | 1.42 |
| > Light the protection or | Atta M Kill on all total |

| Light the archarge: | \$3% pit bill man, ~ 1,000 |
|------------------------|----------------------------|
| COTHER PROMISED FOR | 140 x 1011 (cm//sector) |
| | Che Andre more Page, |
| | meaning at 35° C |
| | fishings (It-Co.Sunge) |
| | metrod |
| Water Conferê | 31% to make 4 in conven |
| | anina. |
| Eurface Write Condent: | 2 80% |

Long Parameter 13.5 to 13.5 cm -20.00 to 120.000 8.5 to 9.2 mm

16.1 mm; 0.134 mm; 40 -0.13401 (pm) 45 4.6 mm; -0.50 m -0.4000 (p.1340 -0.50 m -0.400 (p.1340 -0.50 mm; 6) -0.54 m -0.50 (0.1340 mm; 6)

DAR DES TOTALY 'Adultional features and 'ALROS DARFO trayed

\* Direct Dissertion: 154, 1 acm

\* Contract Dissertion: 154, 1 acm

\* Contract Dissertion: 154, 1 acm

\* Direct Dissertion: 154, 2 acm

\* Direct Contract Dissertion: 154, 2 acm

\* Provers: 49,000 = 140,000

DIMERATIONS (USES)

DIMERATIONS (USES)

DIMERATIONS (USES)

DIMERATIONS (USES)

Reduced for the spiced correction of relución enablegis (1955)

des de hyposofis in hyposofic enables presents with more destruct
popular single probable or apparet presents with more destruct
popular single servicio resultation (O) all assignations flució
core and bendere with whening excito).

DIMERATIONAL "Muddle consideration (O) all assignations flució
core and bendere with whening excito).

DIMERATIONAL "SINGLE SERVICION (O) all assignations flución
portation for the overall convention of remandre annotation place place
and hyposofis resider preschoption is planted in administration of
all conductation for the single confidence as residence plating or
all conductation for the single confidence as residence distinction
and conductation for the single confidence as residence distinction
and conductation for the single confidence and conductation of
all conductations for the single conductation and conductation of
all conductations for the single conductation of
all conductations of the single conductation of
and all conductations of the single conductation of
and conductations of the single conductation of
and conductation of the single conductation of
an all conductations of the single conductation of
an all

displace so to have groundled for ciryle see, shifty dispossible the forces are to be proportion for ciryle see, shifty dispossible sears. The larges are not branched to be observed or distributed and orear. The largest are not inturded to be cloud; be discurded after a pingle gro.

CONTRAINISCRITIONS (PLASONS HOT TO USE)
DO NOT use mideflows & contact linear when any of the
full contraction of contact linear when any of the
full contaction of infection of the mainter chamber of the eye

Active dispass, injury or shearmally stracting the common, originative, or eyeptic the property of the common configuration, or eyeptic the property of the blankwars with control interval property of better the control interval properties of control interval properties of control interval propertie

Problems with cabic lenses and has one probate out read it nations stops to the eye, it is asserted that profess tables their year or protections and stop of their profess tables they are not protected and extended and all high eye between the proper was all phones and since our greatest, afterious pre-probables, helpfulles paramet glowns, can derive profess and limited to be an division. Only one shows are may be detailed all connections and profess about the instruction but to owns fewers wide profess. Of their delivery and the top when that the disk of profess (Device of the processed wine committee) and when the process of the processed wine committee and when the process of the processed wine committee and when the process of the processed wine committee and and the process of the processed of the processed processes. The processed of the processed processes above a triplete includes and others or practices the processes.

recombers.

\*\* I subject to perfector pyr differentiet, burlige budy constitut,
ELECTRIC labels, visit through or reforms of the yet. The
ELECTRIC labels, visit through or reforms of the yet. The
ELECTRIC labels is between the labels of person, became and
party formach is or her eye care protestical, it is
ELECTRIC labels or with the person of the labels of the la

provisional repident as streeted.

PREMATISEES

THE PREMATISEES

THE PREMATISE

THE PREMATISE

THE PREMATISE

THE PREMATISE

THE PREMATISE

THE PREMATISE

THE

by the prescribing any exem professional.

Filamerschia, a pright and quantification is used while the lipease was not the additional open. The limites according to the days and because described the professional open. The control that days and because of the professional open and the control open and the professional open and the company of the professional open and the company of the professional open and the company of

billimet. privile, rijetat receneratis that politicis see their trye core priviletational state each prist, or mere after, as core priviletational state each prist, or mere after, as commonwealthy by the year deep repetitively. District in regimen reduced amonal amounts for their arms prived to core of virgo and on their district see their priviletation of virgo and one priviletation of virgo arms of virg

Eye Cook Professionals should specially indress policies about the following settly presentance:

In following settly presentance:

It a new that before levering the eye term professional a other than professional and the positive the bits promptly resonant below entitled in promptly resonant below entitled in stranger term lesses a finer a demonst also would be a stranger term lesses as the conductable below vower. Always term is, riche and the conductable below vower. Always term is, riche and the conductable below to the conductable belo

But-free Wroal below handling loases,

REMINUS A LINE BARKLINGHEY IF on the sections and of

invitation,

A livery handle lenness carefully, they were to never or other

charp eligible anch as it beyones is to never or other

charp eligible anch as it beyones is to never on the section

they eligible anch as it beyones is to never on the section

to the complete of the section special properties of the section of the

cost level in its never or you because

can level in a never or you because

can level in a never or you because

can level in a never or you have been by as a readired. Since the

cast level in a never or has for an early you is evaluated. Since the

cast level in a never or have been by you in evaluated. Since the

cast level in a never or have been by you in evaluated. Since the

part of the proof to you evaluate properties. I would not be a level or proof of the proof of

Transpromer prometers and the prometer

• While looking sp, alloo to thrue strate man or or mean part of the cpt.
• Remote the love by pictuling partly between the limited and familiar, the next familiar, the next familiar, the next familiar, the next familiar, the press, day frigues cope men to the type of the partle of the specific that is distinct, to great or the partle of the partl

In more occious and marry, it may be payment in recognition.

Claring the days and marry there have the globus, as — Leating in the distriction at the land and disching grant, or — Leating in the distriction at the land and disching grant, or — Court's grant the end of the court in this light disport presence on the adjust of the support of former spike.

If it have been grant and feel and orchordendate, devices were by it is becaused to the organization to the part of an acceleration behind the end of the support of an acceleration behind the end of the support of an acceleration behind the end of the support of an acceleration behind the end of the support of an acceleration behind the end of the support of the end of the support of the end of the support of the end of

Lase Wharing Precediate:

Printed should never crosed the great field unasing schedule
proposition of home constraints the lasess find. Delay as may
increase the claim or constraints the lasess find. Delay as may
increase the claim or should use the age at all deats. If the joint
clotte steps moving in the eye, fallow the recommendate
clottess in the Case also as distingle joint page and
concluses in the Case are as distingle joint joint joint
increases the same that of the place continues, the protocythesis of
includes in the same that of place page continues the protocythesis of
includes the same that they are any contributed of the final continues, the protocythesis of
included to Case and that of place page.

- uri ang lans wakit: kan kacarna dahyeratad ar duruqud. Ca uliti a diadis, kauti, rara lara. Bu carnet lara paner far asah aya la pravani gelisrg
- on agus abus justen angu han as y une pecy-su di agus estas proces angu han as y une pecy-su di agus charactura
- De del mis jeutes jellang gres arbesgan gape.

- To Popule to Oricours with Prillamb?:

  Wholes to Oricours with Prillamb?:

  Wholes the paracticulated are attentionly important he cominate

  can have by Calculus and computed appropriate historia
  control and the paractic state of the paractic historia
  control and the paractic state which year to policial brind sacce

  said year or as recommended by the dynt care protestional,

  contain meadactions are yoursed opposed to the pay, increased

  than eventures, lines beinformer, and illumor brinds or referred

  faccompastions, duration, make relatively, the register, and

  faccompastions, duration, makes relatively, the register, and

  faccompastions, duration, makes relatively, the register, and

  meadactions accordingly and practice proper strengtiff

  meadactions accordingly and practice proper strengtiff

  measures.

he Changed Shows that the Patient is Visoring Contect Learner. Potents and inferent their hardle care presidences that they are a sending remark flower. Foreign model below their enough such that they are wearing contect from the flower that enough such that they are wearing contect from the flower than a content flower and has precident explanation or may require that contact thoses and has precident explanation or may require that contact thoses and has the contact those of the content thoses.

k is stonely recommended that patients to provided with a copy of the BALES TOTALLY and DARRES TOTALLY SARRHOLD Combust Lancest (deliction of ) high oil burdes is small anxieties from Alcon and understand he contents prior to disposaling the lowers.

Appendix expects. Professional to shack eyes regularly to make your tory hand will, and constructed a und without it drive. Principles for the completions are security accomplished by one ay man of the following it gives a propriation.

• Microsia is severe on play any drive of the pro-fession of the following its propriation. — The following is a propriation of the propriation of the pro-fession of the propriation of the propriation of the pro-fession of the propriation of the propriation of the pro-served of the propriation of the propriation of the pro-ter of the propriation of the propriation of the pro-terior polysiscond to the propriation of the propriation of the pro-terior polysiscond to the propriation of the propriation of the pro-terior propriation of the propriation of the propriation of the pro-terior propriation of the propriation of the propriation of the pro-terior propriation of the propriation of the propriation of the pro-terior propriation of the propriation of the propriation of the propriation of the pro-terior propriation of the propriation of the propriation of the propriation of the propriation of the pro-terior propriation of the

- or neutring or other eye secretions richales pulsed discharge

- reggi al 17 a 1704 laghalife fhafa seculificht rinng, singing an hisbing an ansan pais kurani alaad nith Ma
- oyez Combat is how compared to school the lace was first placed an

- I hearing as spinuls occupied.

  Pallent's should be instructed that if may set the altern rights or proposed as the change of proposed are such should.

  I have incoming one produces should be incoming one produced as the change.

  I the alternative one produces alter, notices the first and should be incoming one produces alter, nonevering and the change of the produces on the produces after removing the produces of a new force, Philipping or specific as the produce of a new force, Philipping of the change of the produces of a new force, Philipping of the change of the produces of a new force, Philipping of the produces of the produ
- perfect stands he browned that a perious compiler perfect stands he browned that a perious compiler personal along browned that a perious compiler

ALFORNEE ESFECT REFORMS IN STATES SAFINGE CHICAD RESOLUTION WITH It spellers appealments may reform adoption of the safing and with the case of UNLIES TOTALLY branch desiration is constant inners. Spellers promy, from bracked Sarby in the USA at 1-200-757-6718.

Persia news. Road-Printing String in the USA at L-300-YST-4076.
PITTING CALIDE AND PATISITY DOCURT
Conventional methods of lifeting method houses apply to delinithese A control between Control and Control and the River in the Persia refer to the Control and Control and Control and Control and Control persia and Control and Contr

ASPACIENCY LERES CARE Machig and destruction of dudy at specials innece in ant Consecution. The patient should be remissed in have placement jumes or back-up spectache and table at all divise.

EMERICATES
The product about to informed that if observation of any livel foundation products, greatering collected, foundation products, greatering collected, foundation of any livel foundation of the product of the

| | Spray Spring |
|---|---|
| tree about | |
| 4 | TATE hand in order hand cutter by details in the first order to be by the contract of the cont |
| Jeropa II | Stave do i vel |
| V Da | Life by éta (is pry dest) |
| 1201 | tan wa |
| (3) | Che mad special |
| - 13 | On real area P HE year packages he districted |
| <b>-</b> | Cannyth of test farter forquises code (Crebit) |
| 340 | Chambe |
| #6 | Sun cert |
| PAR | Platf |
| | (Capter Bots presit) |
| ACO | All dan provi |
| (Em | Compani wedwach siçt |
| | CAME |
| rin - | See product rustration |
| | Agricult Representative Services Community |
| | Uplayer |
| | Linguished marge cause 1984 |

4214-1013-149

I Create for estade present mechanism and automoral parameters may be inspected over new term.

I School CO. Chen B.L. Propin BC declare Jin Conyrello. The backer this collection of Control of the backer this propin be a selected from the selected of the propin beautiful propins.

Control deceased, B. Con J. Made. 1868. 27321 (PZ) 773-738.



This page intentionally left blank

This page intentionally left blank

# Alcon

a Novartis company

Manufacturer: Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX 76134-2099, USA

© 2016 Novartis
\*a trademark of Novartis

March 2016

www.alcon.com W900087400-0316

32

# APPENDIX I: CLINICAL TECHNICAL PROCEDURES

- LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS
- EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING
- DETERMINATION OF NEAR ADD
- NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE
- LENS FITTING CHARACTERISTICS
- SUBJECT REPORTED OCULAR SYMPTOMS
- DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS
- BIOMICROSCOPY SCALE
- KERATOMETRY PROCEDURE
- DISTANCE AND NEAR VISUAL ACUITY EVALUATION
- ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE
- MEASURING PUPIL DIAMETER WITH NEUROPTICS VIP-200 VARIABLE PUPILLOMETER

## , LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS
















## **EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING**









# DETERMINATION OF NEAR ADD





























#### LENS FITTING CHARACTERISTICS












### SUBJECT REPORTED OCULAR SYMPTOMS



# DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS
















#### BIOMICROSCOPY SCALE













#### , KERATOMETRY PROCEDURE

5860, v3.0 Amendment 2.0  JJVC CONFIDENTIAL



#### DISTANCE AND NEAR VISUAL ACUITY EVALUATION

5860, v3.0 Amendment 2.0  JJVC CONFIDENTIAL


















# MEASURING PUPIL DIAMETER WITH NEUROPTICS VIP-200 VARIABLE PUPILLOMETER







## PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: <u>CR-5860 Evaluation of Two Marketed Multifocal Contact</u> Lenses

Version and Date: v3.0 Amendment 2.0, 01-SEPT-2017

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to GCP and ICH guidelines, the Declaration of Helsinki, ISO 14155, United States (US) Code of Federal Regulations (CFR), and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution /S't A 11 | |
| | Institution/Site Address | |